

## Clinical Development

# AIN457/ Secukinumab/Cosentyx®

## CAIN457A2323 / NCT02748863

A multicenter, randomized, double-blind, placebocontrolled, 52-weeks study to demonstrate the efficacy, safety and tolerability of subcutaneous secukimumAb injections with 2 mL pre-fiLLed syringes (300 mg) in adUlt subjects with moderate to seveRE plaque psoriasis (ALLURE)

Statistical Analysis Plan (SAP)

Author: Statistician,

stician,

Document type: SAP Documentation

Document status: Addendum 1.0

Release date: 11 Sep 2018

Number of pages: 58

Property of Novartis
For business use only
May not be used, divulged, published or otherwise disclosed
without the consent of Novartis



## **Table of contents**

| | | . Conton | | |
|---|---|---|---|---|
| | Table | e of conte | nts | 3 |
| | List o | of abbrevi | ations | 5 |
| 1 | Intro | duction | | 7 |
| | 1.1 | Study d | lesign | 7 |
| | 1.2 | Study o | objectives and endpoints | 8 |
| 2 | Statis | stical metl | hods | 9 |
| | 2.1 | Data an | nalysis general information | 9 |
| | | 2.1.1 | General definitions | 10 |
| | 2.2 | Analys | is sets | 11 |
| | | 2.2.1 | Subgroup of interest | 12 |
| | 2.3 | Patient | disposition, demographics and other baseline characteristics | 12 |
| | | 2.3.1 | Patient disposition | 13 |
| <ul> <li>Patient disposition, demographics and other baseline characteristics 2.3.1 Patient disposition</li></ul> | | 13 | | |
| | | 2.4.1 | Study treatment / compliance | 13 |
| | | 2.4.2 | Prior, concomitant and post therapies | 16 |
| | 2.5 | Analys | is of the primary objective | 18 |
| | | 2.5.1 | Primary endpoint | 18 |
| | | 2.5.2 | Statistical hypothesis, model, and method of analysis | 22 |
| | | 2.5.3 | Handling of missing values/censoring/discontinuations | 23 |
| | | 2.5.4 | Supportive analyses | 24 |
| | 2.6 | Analysis of the key secondary objective | | |
| | | 2.6.1 | Key secondary endpoint | 24 |
| | | 2.6.2 | Statistical hypothesis, model, and method of analysis | 24 |
| | | 2.6.3 | Handling of missing values/censoring/discontinuations | 25 |
| | 2.7 | Analys | is of secondary efficacy objective(s) | |
| | | 2.7.1 | Secondary endpoints | 25 |
| | | 2.7.2 | Statistical hypothesis, model, and method of analysis | 26 |
| | | 2.7.3 | Handling of missing values/censoring/discontinuations | 26 |
| | 2.8 | Safety a | analyses | 26 |
| | | 2.8.1 | Adverse events (AEs) | 27 |
| | | 2.8.2 | Deaths | 29 |
| | | 2.8.3 | Laboratory data | 29 |
| | | 2.8.4 | Other safety data | 32 |
| | 2.9 | Pharma | acokinetics | 32 |

| | 2.11 | Clinicia | nn-reported outcomes | 33 |
|---|---|---|---|---|
| | | 2.11.1 | Usability and hazard assessment of the 2 mL pre-filled syringe | 33 |
| | 2.12 | Patient- | reported outcomes | 34 |
| | | | | 35 |
| | | | | 35 |
| | | | | 36 |
| 3 | Samp | le size ca | lculation | 36 |
| | 3.1 | Primary | endpoint (co-primary endpoint) | 37 |
| | | 3.1.1 | Secondary endpoints | 37 |
| 4 | Chang | ge to prot | ocol specified analyses | 37 |
| 5 | Appendix | | | |
| | 5.1 | Imputat | ion rules | 37 |
| | | 5.1.1 | Study drug | 37 |
| | | 5.1.2 | AE date imputation | 38 |
| | | 5.1.3 | Concomitant medication date imputation | 39 |
| | | 5.1.4 | First diagnosis date (PsO, PsA) imputation | 40 |
| | | 5.1.5 | Other imputations | 41 |
| | 5.2 | AEs co | ding/grading | 41 |
| | 5.3 | Laborat | ory parameters derivations | 41 |
| | 5.4 | 5.4 Statistical models | | |
| | | 5.4.1 | Analysis of continuous data | 41 |
| | | 5.4.2 | Analysis of binary (and categorical) data | 42 |
| | | 5.4.3 | Logistic regression | 42 |
| | | 5.4.4 | Multiple imputations for response variables | 43 |
| | | 5.4.5 | Crude incidence and related risk estimates | 46 |
| | | 5.4.6 | Exposure adjusted incidence rate and related risk estimates | 48 |
| | 5.5 | Rule of | exclusion criteria of analysis sets | 49 |
| | 5.6 | Clinicia | nn reported outcomes | 49 |
| | | 5.6.1 | Usability and hazard assessment of the 2 mL pre-filled syringe | 49 |
| | 5.7 | Patient | reported outcomes | 51 |
| | | 5.7.1 | Dermatology Life Quality Index (DLQI) | 51 |
| | | | | 52 |
| | | 5.7.3 | Self-injection Assessment Questionnaire (SIAQ) | 54 |
| _ | D C | | | <i></i> |

#### List of abbreviations

AE Adverse event

ALP Alkaline phosphatase

ALT Alanine aminotransferase/glutamic pyruvic transaminase/GPT

AST Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT

ATC Anatomical Therapeutic Chemical

BMI Body Mass Index BSA Body surface area

CHMP Committee for medicinal products for human use

CSR Clinical study report

CTCAE Common Terminology Criteria for Adverse Events

DAR Dosage Administration Record
DLQI Dermatology Life Quality Index

ECG Electrocardiogram

eCRF Electronic case report/record form

FAS Full analysis set

FDA United States Food and Drug Administration

GGT Gamma-glutamyl transferase

HGB Hemoglobin

IFU Instructions For use

IGA Investigator's global assessment

IGA mod 2011 Novartis Investigator's Global Assessment modified 2011

IRT Interactive response technology

LLN Lower Limit of Normal LPLV Last patient's last visit

MACE Major Adverse Cardiovascular Event

MCMC Markov Chain Monte Carlo

MedDRA Medical Dictionary for Regulatory Activities

NMQ Novartis MedDRA Query

NovDTD Novartis Drug and Therapy Dictionary
PASI Psoriasis Area and Severity Index

PD Protocol deviation
PFS Pre-filled syringe
PT Preferred Term

RMP Risk Management Plan

S.C. Subcutaneous

SAS Statistical analysis software SAE Serious adverse event

SIAQ Self-Injection Assessment Questionnaire

SPP Safety Profiling Plan SOC System Organ Class

TBL Total bilirubin

TEAE Treatment Emergent Adverse Event

ULN Upper Limit of Normal

| Novartis | For business use only | Page 6 |
|----------|-----------------------|--------------|
| SAP | | CAIN457A2323 |

WBC White blood cell

## 1 Introduction

Data will be analyzed by Novartis according to the data analysis section 9 of the study protocol which is available in Appendix 16.1.1 of the CSR. Important information is given in the following sections and details are provided, as applicable, in Appendix 16.1.9 of the CSR.

This document covers statistical and analytical plans for CAIN457A2323 (ALLURE) study with reference to the study protocol and the project standard analysis plans (AIN457A Master Analysis Plan).

## 1.1 Study design

This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial in approximately 210 subjects with moderate to severe chronic plaque-type psoriasis.

**Randomization**: Eligible subjects will be randomized using a 1:1:1 ratio into one of the three treatment groups below. Randomization will not be stratified.

- Secukinumab 300 mg (2mL PFS): will receive one 2 mL secukinumab 300 mg plus two 1 mL matching secukinumab placebo s.c. injections once weekly for four weeks (at Randomization, Weeks 1, 2 and 3), followed by dosing every four weeks, starting at Week 4 up to Week 48. Subjects will receive three placebo injections at Weeks 13, 14 and 15.
- Secukinumab 300 mg (2x1mL PFS): will receive two 1 mL secukinumab 150 mg plus one 2 mL matching secukinumab placebo s.c. injections once weekly for four weeks (at Randomization, Weeks 1, 2 and 3), followed by dosing every four weeks, starting at Week 4 up to Week 48. Subjects will receive three placebo injections at Weeks 13, 14 and 15.
- **Placebo**: will receive secukinumab placebo (two 1 mL and one 2 mL s.c. injections) once weekly for four weeks (at Randomization, Weeks 1, 2 and 3), followed by dosing every four weeks, starting at Week 4 up to Week 12 (pre-dose).
  - Prior to receiving the Week 12 dose, all subjects from the **placebo group** will be assigned to the following treatment groups based on their PASI 90 response status as Week 12.
  - PASI 90 non-responders: will receive either one 2 mL 300 mg secukinumab s.c. plus two 1 mL matching placebo OR two 1 mL 150 mg secukinumab s.c. injections plus one 2 mL matching placebo, according to the pre-assignment at the Randomization visit using 1:1 ratio, at Weeks 12, 13, 14, 15 and then every four weeks starting at Week 16 up to Week 48;
  - **PASI 90 responders**: will continue on placebo (one 2 mL plus two 1 mL s.c. injections) and will receive their placebo injections at Weeks 12, 13, 14, 15 and then every four weeks starting at Week 16 up to Week 48.

Of note: For PASI 90 non-responders in **placebo group**, pre-assigned treatment groups at Randomization visit will be used instead of re-randomization at Week 12, therefore eligible subjects will be randomized using pre-assigned 2:2:1:1 ratio into one of the four treatment groups at Randomization visit (similar to 1:1:1 for all subjects at Randomization visit with 1:1 for PASI 90 non-responders in placebo group at Week 12).

• Secukinumab 300 mg (2mL PFS)

- Secukinumab 300 mg (2x1mL PFS)
- Placebo Secukinumab 300 mg (2mL PFS)
- Placebo Secukinumab 300 mg (2x1mL PFS)

The following study periods will be considered for analysis:

- Screening period (before Randomization)
- Treatment period 1 (Randomization to Week 12 pre-dose), including follow-up period (F4 and F8 visits) for prematurely discontinued subjects before Week 12 completion.
- Treatment period 2 (Week 12 dose to Week 52), including follow-up period (F4 and F8 visits) for prematurely discontinued subjects before Week 52 completion.
- Entire treatment period (Randomization to Week 52, last dose at Week 48), including follow-up period (F4 and F8 visits) for prematurely discontinued subjects.

Of note: data from follow-up period (i.e., treatment free follow-up period after EOT visit, which includes F4 and F8 visits) for prematurely discontinued subjects will be included in the analysis of treatment period.

## 1.2 Study objectives and endpoints

The primary objective of this study is to demonstrate the efficacy of secukinumab 300 mg when administered as 2 mL pre-filled syringes in subjects with plaque-type psoriasis with respect to both PASI 75 and IGA mod 2011 0 or 1 response rates at Week 12, compared to placebo.

The key secondary objectives are

- 1) to demonstrate the efficacy of secukinumab 300 mg when administered as 2 mL prefilled syringes versus placebo with respect to:
  - PASI 90 response at Week 12
  - PASI 100 response at Week 12
- 2) to demonstrate the efficacy of secukinumab 300 mg when administered as two 1 mL pre-filled syringes versus placebo with respect to:
  - PASI 100 response at Week 12

Furthermore, additional aspects of efficacy, safety and tolerability of secukinumab 300 mg as 2 mL pre-filled syringes compared to secukinumab 300 mg as two 1 mL pre-filled syringes over a period of 52 weeks will be investigated.

This study will provide efficacy and safety data to support a product labeling updates for the indication of moderate to severe plaque psoriasis.

Table 1-1 Primary, key secondary, secondary and exploratory variables

| | Туре |
|--------------------------------------------------|---------------|
| PASI 75 response @ Week 12 | primary |
| IGA 0/1 response @ Week 12 | primary |
| PASI 90 response @ Week 12 | key secondary |
| PASI 100 response @ Week 12 | key secondary |
| PASI 50/75/90/100 and IGA 0/1 response over time | secondary |
| PASI score and IGA mod 2011 categories over time | secondary |
| Device usability (IFU and use-related hazards) | secondary |
| SIAQ | secondary |
| DLQI score | secondary |
| DLQI 0 or 1 achievement | secondary |
| DEQL 0 or 1 achievement | secondary |

## 2 Statistical methods

## 2.1 Data analysis general information

| Novartis will be performing final | analysis. | Statistical |
|-------------------------------------------------|-----------|-------------|
| software SAS version 9.4 or later will be used. | | |

Summary statistics for continuous variables will include N, mean, standard deviation, minimum, lower quartile, median, upper quartile, maximum. Summary statistics for discrete variables will be presented in contingency tables and will include absolute and relative frequencies.

The p-values will be presented as one-sided for hypothesis testings and as two-sided for other analysis. Two-sided 95% confidence intervals will be displayed. If not otherwise specified, hypothesis testings will be based on one-sided p-values that the treatment effect is in favor of Secukinumab. The level of significance will be set to 2.5% (one-sided, family-wise type-I-error). The 95% confidence intervals will not be used for decision making; they will only be used for estimation and will therefore always be two-sided.

All listings will be presented by treatment sequence.

Footnotes on outputs will be kept to a minimum also for outputs not covered in [MAP TFL shells].

Footnotes will generally be provided for

• abbreviations used in the output; abbreviations used on several outputs, e.g. for listings in Appendix 16.2 can be presented on a separate page and do not have to be repeated as footnotes on each listing

- sorting order of categories, e.g. for sorting within MedDRA (Medical Dictionary for Regulatory Activities) hierarchy levels
- MedDRA version used for reporting of MedDRA coded data

Footnotes will generally NOT be given for

- units displayed on the output
- interpretation of results (e.g. "odds ratio larger than 1 favors active treatment")
- information that can be retrieved from the statistical section of the clinical study report (CSR) unless it is not identifiable from the output, e.g.
  - explanation of analysis model used unless results of more than one model are displayed on an output
  - derivations of variables (e.g. BMI will not be explained on a footnote)
- information that will be provided in the clinical study protocol and/or methods section of the CSR (e.g. baseline definition if this is specified in the statistical section of the CSR)

#### 2.1.1 General definitions

## 2.1.1.1 Study treatment

The following study drugs will be used:

- Investigational treatment
  - o Secukinumab 300 mg, 2 mL liquid formulation in a pre-filled syringe
- Control treatment
  - o Secukinumab 150 mg, 1 mL liquid formulation in a pre-filled syringe
  - o Secukinumab placebo, 2 mL liquid formulation in a pre-filled syringe
  - o Secukinumab placebo, 1 mL liquid formulation in a pre-filled syringe

#### 2.1.1.2 Study Day 1 and other study days

The first day of administration of randomized study treatment (first dose) is defined as *Study Day 1* or *Day 1*.

All other study days will be labeled relative to Day 1. For event dates on or after Day 1, study day for a particular event date is calculated as [Date of event] – [Date of first dose]+1, i.e., Day 2, Day 3, etc., will be one day, two days, etc., after Day 1, respectively. For the dates before Day 1, study day for an event date is calculated as [Date of event] – [Date of first dose], i.e., Day -1, Day -2, etc., will be one day, two days, etc., before Day 1, respectively. Duration of an event will be calculated as (Event end date – Event start date + 1).

The descriptor "Day 0" will not be used.

#### 2.1.1.3 Screening, baseline and post-baseline definitions

Screening refers to any procedures (e.g., checking inclusion and exclusion criteria) performed prior to the date of first dose of study treatment (for safety analysis) or prior to the randomization

date (for efficacy analysis). Per protocol, subject informed consent must be obtained prior to performing any study related activity. The date of signing informed consent is the start date of screening period. Any assessment obtained during the screening period will be labeled screening assessment. Assessments made on Day 1 may occur before or after the randomization or the first dose.

For <u>efficacy</u> analyses, baseline is the last assessment (including unscheduled visits) obtained (on or) before the randomization (day). All assessments obtained after randomization (day) are considered as post-baseline unless otherwise specified.

For <u>safety</u> analyses, baseline is the last assessment (including unscheduled visits) obtained (on or) before the first dose (day) of study treatment. All assessments obtained after the first dose (day) of study treatment are considered as post-baseline unless otherwise specified.

In general, a baseline value refers to the last measurement made prior to administration of the first dose of study treatment. However, for PROs, LAB assessments and ECG if no pretreatment value exists, values obtained after first dose of treatment can be used as baseline <u>only</u> if it was collected on the same day as first dose.

## 2.1.1.4 Day of last dose of randomized study treatment

The date of last dose will be collected via the CRF.

Duration of exposure is defined in Section 2.4.1.

On-treatment is defined as assessments within last dose plus 84 days.

## 2.2 Analysis sets

The following analysis sets will be used for the data analysis.

**Randomized set:** The randomized set will be defined as all subjects who were randomized at baseline visit. Unless otherwise specified, mis-randomized subjects will be excluded from the randomized set.

Misrandomized subjects are subjects who are screen-failures, but have been randomized by the investigator before eligibility was finally assessed, however have not been treated. If previously mis-randomized subjects were re-screened and successfully randomized, they will be included in the randomized set according to the treatment assigned in the last randomization.

**Full analysis set (FAS)**: The FAS will be comprised of all subjects from the randomized set to whom study treatment has been assigned. Following the intent-to-treat principle, subjects will be analyzed according to the treatment assigned to at randomization. If the actual randomization stratum is different to the assigned stratum in IRT, the actual stratum will be used in analyses.

Of note, subjects excluded from the randomized set will be excluded from the FAS.

**Safety set**: The safety set includes all subjects who took at least one dose of study treatment during the treatment period. Subjects will be analyzed according to treatment received.

The treatment received will be set to the treatment randomized. But if a subject has received the wrong treatment during the entire study, the treatment received will be set to this wrong treatment.

For those subjects who received erroneously the wrong treatment at least once, an additional listing will be prepared displaying adverse events occurred after the treatment errors.

### 2.2.1 Subgroup of interest

Not applicable.

# 2.3 Patient disposition, demographics and other baseline characteristics

The summaries will be shown for the following treatment groups, before or at Week 12:

- AIN457 300 mg (2mL PFS), AIN457 300 mg (2x1mL PFS), Placebo, Total after Week 12:
- AIN457 300 mg (2mL PFS), AIN457 300 mg (2x1mL PFS), Placebo, Placebo AIN457 300 mg (2mL PFS), Placebo AIN457 300 mg (2x1mL PFS), Total
   No summaries for entire treatment period will be provided.

The following common background and demographic variables will be analyzed:

#### **Continuous variables:**

- Age (which is derived from year of birth and the Informed consent date, assuming date is July 1<sup>st</sup> since only year of birth is collected)
- o Height
- o Weight
- o Body mass index (BMI)

#### Categorical variables:

- o Age categories (<65 years, 65 years and older, 75 years and older)
- o Sex
- o Race
- o Ethnicity
- o Smoking status at baseline

Psoriasis specific baseline characteristics and history of disease will be summarized as well: baseline PASI, baseline PASI ( $\leq 20, > 20$ ), baseline total BSA, baseline IGA mod 2011 score (at least mild, moderate, severe), severity of psoriasis (CHMP guidelines, mild (total BSA  $\leq 10\%$  and PASI  $\leq 10$ ), moderate ((PASI  $\geq 10$  or total BSA  $\geq 10\%$ ) and PASI  $\leq 20$  and total BSA  $\leq 20\%$ ), severe (total BSA  $\geq 20\%$  or PASI  $\geq 20$ )), psoriatic arthritis (yes, no), time since diagnosis of psoriasis, time since diagnosis of psoriatic arthritis, previous exposure to biologic systemic psoriasis therapy, previous exposure to systemic psoriasis therapy, previous exposure to non-biologic systemic psoriasis therapy, previous failure to systemic psoriasis therapy, previous failure to non-biologic systemic psoriasis therapy (including phototherapy and photo-chemotherapy)

Body Mass Index (BMI) will be calculated using the following formula:

 $BMI = (body weight in kilograms) / (height in meters)^2$ 

For BMI, height and body weight the last value prior to randomization is used. If there is no weight recorded prior to taking of study treatment, BMI will be missing.

Of note: subject's height will not be remapped according to the analysis visit window.

Time since diagnosis of psoriasis (PsO) and time since diagnosis of psoriatic arthritis (PsA) will be calculated using the following formula:

Time since diagnosis = (inform consent date - first diagnosis date + 1)/365.25

The first diagnosis date of PsO or PsA will be imputed according to the imputation rules in Section 5.1.

Unless otherwise specified, summary statistics will be presented for continuous variables for each treatment group and for all subjects (total) in the randomized set. The number and percentage of subjects in each category will be presented for categorical variables for each treatment group and all subjects (total) in the randomized set.

Any condition entered on the *relevant medical history / current medical conditions* CRF (including family history) will be coded using the MedDRA dictionary. They will be summarized by System Organ Class (SOC) and Preferred Term (PT) of the MedDRA dictionary.

Summaries for cardiovascular medical history will be summarized by categories.

Smoking history will be summarized by treatment group.

Unless otherwise specified, analyses will be based on the randomized set.

## 2.3.1 Patient disposition

The number of subjects screened will be presented. In addition, the reasons for screen failures will be provided. The number and percentage of subjects in the randomized set who completed study periods and who discontinued the study prematurely (including the reason for discontinuation) will be presented for each treatment group and all subjects.

For each protocol deviation, the number and percentage of subjects for whom the deviation applies will be tabulated.

# 2.4 Treatments (study treatment, concomitant therapies, compliance)

#### 2.4.1 Study treatment / compliance

The analysis of study treatment data will be based on the safety set.

The number of secukinumab 2mL syringes, 1mL secukinumab syringe, secukinumab placebo injections will be summarized by treatment group by means of contingency tables.

The duration of exposure to study treatment will be summarized by treatment group. In addition, the number of subjects with exposure of at least certain time thresholds will be displayed. The following categories will be presented: "any exposure", " $\geq$ 1 week", " $\geq$ 2 week", " $\geq$ 4 weeks", " $\geq$ 8 weeks", " $\geq$ 12 weeks", " $\geq$ 16 weeks", " $\geq$ 28 weeks", " $\geq$ 40 weeks" and " $\geq$ 52 weeks".

Duration of exposure will be defined as the time from first dose of study medication to the last dose plus 84 days or last visit (including follow-up visits) whichever occurs earlier. i.e., for subjects who discontinued or have their last visit earlier than 84 days, the end of study treatment exposure will be the date of the last study visit in the follow-up period or in the corresponding treatment period.

Duration of exposure (days) = min (last study visit (including follow-up) date, last dose date +84) – first dose date +1

Duration of exposure (years) = duration of exposure (days) / 365.25

Duration of exposure (100 subject years) = duration of exposure (years) / 100

#### 2.4.1.1 Visit window

*Visit-windows* will be used for the data that is summarized by visit; they are based on the study evaluation schedule and comprise a set of days around the nominal visit day. For any assessment, there are the protocol defined scheduled visits around which visit windows were created to cover the complete range of days within the study. The visit windows are shown in Table 2-1. In this table, the days are counted since the first dose of study treatment ( Day 1) for safety assessments, and the days are counted since the date of randomization for efficacy assessments. These visit windows apply to measurements taken at every visit.

When visit windows are used, all visits will be re-aligned, i.e., they will be mapped into one of the visit windows. E.g., if the *Week 4* visit of a subject is delayed and occurs on Day 60 instead of on Day 29, it will be re-aligned to visit window *Week 8*. In the case of major deviations from the visit schedule, or due to unscheduled visits, several assessments of a subject may fall in a particular visit window (either scheduled or unscheduled). Statistical approaches to handle multiple assessments in a given visit window are specified below.

For parameters which are not collected at every visit (e.g., DLQI), visit windows will be combined. For example, if a parameter is measured at Week 12 and Week 28 only, Week 12 visit window will extend from Day 2 to Day 99 (combining Week 1 to Week 12 visit windows), and Week 28 will be extend from Day 100 to Day 239.

Assessments from treatment period 2 will not be considered for treatment period 1, and treatment period 1 visits will not be mapped into treatment period 2.

Of note: for subjects who prematurely discontinued, efficacy measurements taken in follow-up period will be remapped to treatment periods.

Table 2-1 Assessment windows for scheduled visits

| Analysis Visit | Week | Scheduled Day | Visit Window |
|----------------|------|---------------|--------------------|
| Baseline | BSL | 1 | -28 days to Day 1* |
| Week 1 | 1 | 8 | Day 2-11 |
| Week 2 | 2 | 15 | Day 12-18 |
| Week 3 | 3 | 22 | Day 19-25 |
| Week 4 | 4 | 29 | Day 26-43 |
| Week 8 | 8 | 57 | Day 44-71 |
| Week 12 | 12 | 85 | Day 72-99 |
| Week 16 | 16 | 113 | Day 100-155 |
| Week 28 | 28 | 197 | Day 156-239 |
| Week 40 | 40 | 281 | Day 240-323 |
| Week 52 | 52 | 365 | Day 324-421 |

<sup>\*</sup> Baseline measurement before the first drug administration for safety assessments and before the randomization for efficacy assessments.

Of note: subject's height will not be remapped according to the analysis visit window.

The analysis visit will be used for listing of visit and period for safety data. If a visit falls after the last visit window (after Day 421) it is not assigned an analysis visit and will be listed under label "After Week 52".

### 2.4.1.2 Multiple assessments within visit windows

When there are *multiple assessments* in a particular visit window, the following rules are applied to select one value "representing" the subject in summary statistics in a visit window (See Table 2-2).

For baseline assessment definition see Section 2.1.1.3. For post-baseline visit windows the following applies (unless otherwise specified):

- for *quantitative variables*, the *closest* to the actual visit is chosen (if two assessments have the same distance, then the earlier one will be chosen);
- for *qualitative variables*, the *worst* record is selected. It is noted that in the analyses performed, *worst* case is always well defined (e.g., for urine protein values "+" and "++", the worst case is defined as "++"),
- in case qualitative variables are based on quantitative variables, e.g. PASI 90 response, the visit will be assigned to the quantitative variable, and this visit will be used for the derived qualitative variable.

Table 2-2 Rules for selecting values for analysis within a given visit window

| Timing of measurement | Type of data | Rule |
|---|---|---|
| Baseline | All data | See Section 2.1.1.3. |
| Post-baseline efficacy | All data except for PRO, e.g., PASI, IGA | The measurement closest to the target day will be used. In the event two measurements are taken equally apart (e.g., 1 day before target date and 1 day after), the earlier one will be used. |
| | | If two measurements are taken on the same day then select the first one using eCRF visit number. |
| | | If two measurements have been taken on the same day and same visit then select the worst. |
| Post-baseline efficacy | PRO data | The measurement closest to the target day will be used. In the event two measurements are taken equally apart (e.g., 1 day before target date and 1 day after), the earlier one will be used. |
| | | If two measurements have been taken on the same day, select the worst. |
| | | If two measurements have the same value, select the first one using eCRF visit number. |
| Post-baseline safety | Summary visit information (e.g. laboratory values, vital signs, etc.) | The (non-missing) measurement closest to the target day will be used. In the event two measurements are taken equally apart (e.g., 1 day before target date and 1 day after), the earlier one will be used. If two measurements are taken on the |
| | | same day then select the first one (using the time). |
| | | If two measurements are taken on the same date/time then use the first eCRF visit number (assuming this is the planned visit). If two measurements are taken on the same date/time/eCRF visit number then take the average value of these two results. |
| Post-baseline safety | Notable abnormalities (e.g. vitals signs) and CTCAE grades for laboratory values | The most extreme measurement in the window will be used. Note this means a subject can have a notably high and notably low measurement within an analysis period. |

## 2.4.2 Prior, concomitant and post therapies

Medications will be identified using Novartis Drug and Therapy Dictionary (NovDTD) including Anatomical Therapeutic Chemical (ATC) code. Prior and concomitant treatments will be summarized by treatment group for the safety set unless otherwise specified. Concomitant treatments will be displayed for the treatment period 1 and entire treatment period.

Prior and concomitant medications will be summarized by treatment group in separate tables. Medications will be presented in alphabetical order, by ATC codes and grouped by *anatomical main group* (the 1<sup>st</sup> level of the ATC codes). Tables will also show the overall number and percentage of subjects receiving at least one drug of a particular ATC code and at least one drug in a particular anatomical main group.

Prior medications are defined as drugs taken and stopped prior to the first dose of study treatment. Any medication given at least once between the day of first dose of randomized study treatment, and last dose plus 84 days or last visit (including follow-up visits) whichever occurs earlier will be a **concomitant** medication, including those which were started pre-baseline and continued into the treatment period.

Summaries of prior and/or concomitant psoriasis specific medication will be presented as in Table 2-3, but as well for topical, phototherapy and photochemotherapy (yes/no) using the randomized set.

In addition, medical procedures and significant non-drug therapies as coded in MedDRA will be summarized.

Prior or concomitant medication will be identified based on recorded or imputed start and end dates of medication taken. Further rules will be given in Section 5.

Table 2-3 Subgroups based on the previous psoriasis therapy

| Level 1<br>description | Level 1 outcome | Level 2 description | Level 2 outcome | Level 3 description | Level 3 outcome | Level 4 description | Level 4 outcome |
|---|---|---|---|---|---|---|---|
| previous<br>therapy | yes/no | | | | | | |
| systemic | no | | | | | | |
| | yes | number | 1 | | | | |
| | | | 2 | | | | |
| | | | >=3 | | | | |
| | | failure* | no | | | | |
| | | | yes | | | | |
| biologic | no | | _ | | | | |
| | yes | failure* | no | | | | |
| | | | yes | | | | |
| | | type of previous | type of previous biologic | | | | |
| | | anti-p40 | no | no | | | |
| | | | yes | failure* | no | | |
| | | | | | yes | | |
| | | anti-TNF | no | T | 1 | | |
| | | | yes | failure* | no | T | T |
| | | | | | effica<br>lack of<br>effica | lack of primary | no |
| | | | | | | | yes |
| | | | | | | lack of secondary | no |
| | | | | | | | yes |
| | | | | | | lack of primary or | no |
| | | | | | | secondary efficacy | yes |
| | | | | | | lack of tolerability | no |
| | | | | | | | yes |
| non-biologic | no | <u> </u> | 1 | | | | |
| systemic | yes | failure* | no | | | | |
| | | | yes | | | | |
| | | failure* to at | no | | | | |
| | | least 2 | yes | | | | |

only selected subgroups will be used for reporting

## 2.5 Analysis of the primary objective

## 2.5.1 Primary endpoint

The co-primary endpoints are PASI 75 response and IGA 0 or 1 response at Week 12. The analysis of the primary variables will be based on the FAS.

#### 2.5.1.1 Definition of PASI and related variables

The investigator or trained qualified designee will complete the PASI assessments. Whenever possible, the same evaluator should perform this assessment at all visits.

The total BSA affected by plaque-type psoriasis will be estimated from the percentages of areas affected, including head, trunk, upper limbs and lower limbs (see below for PASI assessment). The following calculations will be done: each reported percentage will be multiplied by its respective body region corresponding factor (head = 0.1, trunk = 0.3, upper limbs = 0.2, lower

<sup>\*:</sup> at least one therapy with lack of primary efficacy or lack of secondary efficacy or lack of tolerability

limbs = 0.4). The resulting 4 percentages will be added up to estimate the total BSA affected by plaque-type psoriasis. The PASI scoring system is further described in Table 2-4.

A PASI score (Fredriksson and Pettersson 1978, Weisman et al 2003, Gottlieb et al 2005) will be derived as indicated in Table 2-4. The head, trunk, upper limbs and lower limbs are assessed separately for erythema, thickening (plaque elevation, induration), and scaling (desquamation). The average degree of severity of each sign in each of the four body regions is assigned a score of 0-4. The area covered by lesions on each body region is estimated as a percentage of the total area of that particular body region. Further practical details help the assessment:

- 1. The neck is assessed as part of the head.
- 2. The axillae and groin are assessed as part of the trunk.
- 3. The buttocks are assessed as part of the lower limbs.
- 4. When scoring the severity of erythema, scales should not be removed.

Because the head and neck, upper limbs, trunk and lower limbs correspond to approximately 10%, 20%, 30% and 40% of the body surface area, respectively, the PASI score will be calculated using the formula:

$$PASI = 0.1 (E_h + I_h + D_h)A_h + 0.2 (E_u + I_u + D_u)A_u + 0.3 (E_t + I_t + D_t)A_t + 0.4 (E_l + I_l + D_l)A_l$$

where E, I, D, and A denote erythema, induration, desquamation, and area, respectively, and h, u, t, and l denote head, upper extremities, trunk, and lower extremities, respectively (see Table 2-4).

PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0.

The investigator is responsible for collecting the components or scoring signs and total regional area for all visits. Total PASI and total BSA calculations will be done by investigator at screening and randomization only; The total PASI and BSA scores will be calculated by Novartis and will be used in the analysis and for derivation of PASI response values (see below).

Table 2-4 The PASI scoring system

| Body<br>region | Erythema (E) | Thickening<br>(plaque elevation,<br>induration, l) | Scaling<br>(desquamation,<br>D) | Area score<br>(based on true<br>area %, A)* |
|---|---|---|---|---|
| Head (H) <sup>†</sup> | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0 = no involvement<br>1 = >0-<10%<br>2 = 10-<30%<br>3 = 30-<50%<br>4 = 50-<70%<br>5 = 70-<90%<br>6 = 90-100% |
| Trunk (T) <sup>‡</sup> | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0 = no involvement<br>1 = >0-<10%<br>2 = 10-<30%<br>3 = 30-<50%<br>4 = 50-<70%<br>5 = 70-<90%<br>6 = 90-100% |
| Upper<br>limbs (U) | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0 = no involvement<br>1 = >0-<10%<br>2 = 10-<30%<br>3 = 30-<50%<br>4 = 50-<70%<br>5 = 70-<90%<br>6 = 90-100% |
| Lower<br>limbs (L)§ | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0=none<br>1=slight<br>2=moderate<br>3=severe<br>4=very severe | 0 = no involvement<br>1 = >0-<10%<br>2 = 10-<30%<br>3 = 30-<50%<br>4 = 50-<70%<br>5 = 70-<90%<br>6 = 90-100% |

<sup>\*</sup> Percentage (not score) of body region (not whole body) affected will be entered in the eCRF.

The following definitions are possible efficacy evaluations that can be used in clinical trials in psoriasis (CHMP/EWP/2454/02, 2004):

- **PASI 50 response**: subjects achieving ≥ 50% improvement (reduction) in PASI score compared to baseline are defined as PASI 50 responders
- **PASI 75 response**: subjects achieving ≥ 75% improvement (reduction) in PASI score compared to baseline are defined as PASI 75 responders
- **PASI 90 response**: subjects achieving ≥ 90% improvement (reduction) in PASI score compared to baseline are defined as PASI 90 responders
- PASI 100 response / remission: complete clearing of psoriasis (PASI=0)

<sup>&</sup>lt;sup>†</sup> Neck is assessed as part of the Head (H) body region.

<sup>&</sup>lt;sup>‡</sup> Axillae and groin are assessed as part of the Trunk (T) body region.

<sup>§</sup> Buttocks are assessed as part of the Lower limbs (L) body region.



## 2.5.1.2 Definition of IGA mod 2011 score and IGA mod 2011 0 or 1 response

The IGA mod 2011 rating scale for overall psoriatic disease (shown in Table 2-5) has been developed based on a previous version of the scale used in secukinumab phase II studies, and has been updated in collaboration with health authorities (in particular the FDA). The explanations/descriptions of the points on the scale have been improved to ensure appropriate differentiation between the points. It is recommended that the same evaluator conducts the assessments throughout the study whenever possible.

The IGA mod 2011 used in this study is static, i.e., it refers exclusively to the subject's disease state at the time of the assessments, and does not attempt a comparison with any of the subject's previous disease states, whether at baseline or at a previous visit.

Table 2-5 The IGA mod 2011 rating scale

| Score | Short Description | Detailed Description |
|---|---|---|
| 0 | Clear | No signs of psoriasis. Post-inflammatory hyperpigmentation may be present. |
| 1 | Almost clear | Normal to pink coloration of lesions; no thickening; no to minimal focal scaling. |
| 2 | Mild | Pink to light red coloration; just detectable to mild thickening; predominantly fine scaling. |
| 3 | Moderate | Dull bright red, clearly distinguishable erythema; clearly distinguishable to moderate thickening; moderate scaling. |
| 4 | Severe | Bright to deep dark red coloration; severe thickening with hard edges; severe / coarse scaling covering almost all or all lesions. |

Note: Involvement of nails is not part of the assessment.

Subjects require an IGA mod 2011 score at randomization of 3 or 4 in order to participate in the study. Based on this scale, subjects will be considered as **IGA mod 2011 0 or 1 responder** if they achieve a score of 0 or 1 and improve by at least 2 points on the IGA mod 2011 scale compared to baseline.

#### 2.5.1.3 Overview of analysis methods of efficacy variables

An overview of statistical analyses and methods applied to psoriasis efficacy variables is given in Table 2-6.

Table 2-6 Overview of analysis methods for efficacy variables

| Variable(s) | Summary<br>statistics for<br>binary/<br>categorical data | Logistic regression | Summary<br>statistics for<br>continuous<br>data | Time-to-<br>event<br>analysis | Graphs |
|---|---|---|---|---|---|
| PASI 75 response @ Week 12 | Х | Х | | | X* |
| IGA 0/1 response @ Week 12 | Х | X | | | X* |
| PASI 90 response @ Week 12 | Х | X | | | X* |
| PASI 100 response @ Week 12 | Х | X | | | X* |
| PASI 50/75/90/100 and IGA 0/1 response over time | Х | Х | | | X** |
| PASI score over time | | | Х | | X** |
| IGA mod 2011 categories over time | Х | | | | |
| Device usability (IFU and use-related hazards) | Х | | | | |
| SIAQ | | | Х | | |
| DLQI score over time | | | Х | | |
| DLQI 0/1 over time | Х | | | | |
| * dot plot; ** time course plot | | | | | |

## 2.5.2 Statistical hypothesis, model, and method of analysis

The statistical hypotheses are that secukinumab 300 mg (2mL PFS) is not superior to placebo in the proportion of subjects with PASI 75 response and IGA 0 or 1 response at Week 12.

Let  $p_j$  denote the proportion of PASI 75 responders at Week 12 for treatment group j and  $r_j$  denote the proportion of IGA 0 or 1 responders at Week 12 for treatment group j;

j=0, 1, where

- 0 corresponds to placebo,
- 1 corresponds to secukinumab 300 mg (2mL PFS).

The following hypotheses will be tested:

H:  $H_1 \cup H_2$  versus  $H_A$ :  $H_{A1} \cap H_{A2}$ 

 $H_1$ :  $p_1 - p_0 \le 0$  versus  $H_{A1}$ :  $p_1 - p_0 \ge 0$ ,

 $H_2$ :  $r_1 - r_0 \le 0$  versus  $H_{A2}$ :  $r_1 - r_0 \ge 0$ 

In other words:

H: secukinumab 300 mg (2mL PFS) is not superior to placebo with respect to either PASI 75 response at Week 12 or IGA 0 or 1 response at Week 12 or both

H<sub>1</sub>: secukinumab 300 mg (2mL PFS) is not superior to placebo with respect to PASI 75 response at Week 12

H<sub>2</sub>: secukinumab 300 mg (2mL PFS) is not superior to placebo with respect to IGA 0 or 1 response at Week 12

The primary analysis method for PASI 75 and IGA 0 or 1 response at Week 12 will be evaluated using logistic regression model with treatment group, baseline bodyweight and baseline PASI score as explanatory variables (see Section 5 Appendix). Odds ratios will be computed for

comparisons of secukinumab dose regimen versus placebo utilizing the logistic regression model fitted. In case of the logistic regression does not converge due to low response rates in the placebo group, an exact logistic regression will be performed. In case of response rates of 0% or 100% in one of the treatment groups, for analyses with multiple imputation, confidence intervals for risk difference and p-values from the t-test for the risk difference comparing to 0 will be provided; for analyses with non-responder imputation, Fisher's exact test will be performed and confidence intervals for risk difference will be provided.

The hypotheses  $H_1$  and  $H_2$  will both be tested at  $\alpha$  level = 2.5% (one-sided) and significant results will only be achieved if both hypotheses are rejected (i.e., if only one hypothesis is rejected and the other hypothesis is not rejected, superiority of secukinumab 300 mg 2mL PFS cannot be demonstrated).

The primary analysis set will be the FAS.

Summary statistics and figures will be provided as described in Section 5.4.2. Details in sensitivity analysis are provided in Section 2.5.4.

## 2.5.3 Handling of missing values/censoring/discontinuations

Response variables based on PASI score and IGA mod 2011 categories will be imputed with multiple imputation (MI) as primary imputation method for the missing values.

Multiple imputation (MI) is a simulation based approach where missing values are replaced by multiple Bayesian draws from the conditional distribution of missing data given the observed data and covariates, creating multiple completed data sets. These completed data sets can then be analyzed using standard methods. Within this analysis the PASI score or IGA mod 2011 categories will be imputed and response variables will be derived based on the imputed scores. In the multiple imputation analysis the response status will be imputed based on the individual treatment arm information.

(Modified) Non-responder imputation will be used as a sensitivity method: Missing values with respect to response variables based on PASI score and IGA 2011 categories will be imputed with non-response regardless to the reason for missing data (e.g. premature study discontinuation, missed visit, administrative issues), exceptions will apply to the following:

- If a subject dropped out of the study prior to last scheduled visit and being responder consecutively at least for two preceding visits before drop-off, the subject will be imputed as responder for all the later visits till last scheduled visit.
- If a subject who was responder at visit *x*-1 and visit *x*+1 but has missing data at visit *x*, then the subject will be imputed as responder for visit *x* as long as the distance between the scheduled visits *x*-1 and *x* is 4 weeks or less, and the distance between the scheduled visits *x* and *x*+1 is 4 weeks or less. Otherwise missing data will be imputed with non-response.

Summary tables for PASI scores and IGA mod 2011 categories will be imputed using MI. The mean for PASI score and the number (%) for IGA mod 2011 categories as well as their 95% confidence intervals will be given. In addition, PASI scores and IGA mod 2011 categories based on LOCF imputation will be provided in summary tables and listings.

Note: Only PASI and IGA mod 2011 based response variables are imputed with multiple imputation or non-response, other response variables (e.g. DLQI 0 or 1 achievement) will be imputed with LOCF.

#### 2.5.4 Supportive analyses

Sensitivity analyses will be performed as follows:

(A) Co-primary endpoints (PASI 75 and IGA 0 or 1 response at Week 12) and key secondary endpoints will be evaluated using the logistic regression as described in primary analysis method with non-responder imputations instead of multiple imputation for missing values.

## 2.6 Analysis of the key secondary objective

## 2.6.1 Key secondary endpoint

The key secondary endpoints of this study are planned as follow:

- PASI 90 response at Week 12
- PASI 100 response at Week 12

The null hypotheses for secondary objectives are as follows:

- H<sub>3</sub>: secukinumab 300 mg (2mL PFS) is not superior to placebo with respect to PASI 90 response at Week 12
- H<sub>4</sub>: secukinumab 300 mg (2mL PFS) is not superior to placebo with respect to PASI 100 response at Week 12
- H<sub>5</sub>: secukinumab 300 mg (2x1mL PFS) is not superior to placebo with respect to PASI 100 response at Week 12

#### 2.6.2 Statistical hypothesis, model, and method of analysis

The following hypotheses will be tested sequentially and are included in the hierarchical testing strategy and type-I-error will be set such that a family-wise type-I-error of  $\alpha = 2.5\%$  (one-sided) is kept. The graphical approach of (Bretz et al. 2009) for sequentially rejective testing procedures is used to illustrate the testing strategy:

Figure 1-1 Testing strategy



The secondary efficacy variables involved in the above testing strategy will be analyzed analogously to the primary endpoints. i.e., logistic regression model with treatment group, baseline bodyweight, and baseline PASI score as explanatory variables. Odds ratios will be computed for comparisons of secukinumab regimen versus placebo utilizing the logistic regression model fitted.

The testing sequence will continue to  $H_3$  at  $\alpha$  (one-sided) only if both  $H_1$  and  $H_2$  have been rejected at  $\alpha$  (one-sided). Similarly, the testing sequence will continue to  $H_4$  at  $\alpha$  (one-sided) only if  $H_3$  testing has been rejected. In case,  $H_4$  has been rejected at  $\alpha$  (one-sided), the corresponding alpha ( $\alpha$ ) will be passed to the next hypotheses corresponding  $H_5$ .

#### 2.6.3 Handling of missing values/censoring/discontinuations

See Section 2.5.3.

## 2.7 Analysis of secondary efficacy objective(s)

#### 2.7.1 Secondary endpoints

# PASI 50, PASI 75, PASI 90, PASI 100, and IGA mod 2011 0 or 1 response over time

Summary statistics for PASI 50, PASI 75, PASI 90, PASI 100, and IGA mod 2011 0 or 1 response by visit will be presented in contingency tables and will include absolute and relative frequencies. Confidence intervals for response rates will be derived as well based on the score method including continuity correction (Newcombe 1998).

For PASI 50, PASI 75, PASI 90, PASI 100, and IGA mod 2011 0 or 1 response at each visit, up to Week 12, secukinumab dose regimen will be compared to placebo by means of logistic regression model with treatment group, baseline bodyweight and baseline PASI as effects.

For PASI 50, PASI 75, PASI 90, PASI 100, and IGA mod 2011 0 or 1 response, the placebo adjusted response rates (i.e., risk difference) including 95% confidence interval (based on normal approximation) will be derived by visit, up to Week 12. In addition, Fisher's exact test

will be applied to the treatment group comparisons between secukinumab dose regimens versus placebo.

Figures will be provided for PASI 50, PASI 75, PASI 90, PASI 100, and IGA mod 2011 0 or 1 response over time, by displaying estimates for response rates by treatment including 95% confidence intervals.

## PASI score and IGA mod 2011 categories over time

Summary statistics will be provided for absolute PASI scores and IGA mod 2011 categories, as well as for percentage change from baseline for PASI scores by visit and treatment group. Figure will be provided for percentage changes in PASI scores over time.

#### 2.7.2 Statistical hypothesis, model, and method of analysis

Not applicable.

## 2.7.3 Handling of missing values/censoring/discontinuations

See Section 2.5.3.

## 2.8 Safety analyses

All safety analyses will be based on the safety set. Only those scheduled visits which were preplanned in the protocol will be reported in tables and figures for safety variables.

## Treatment groups for evaluation of entire treatment

The summaries of evaluation will be reported for treatment period 1 and entire treatment period, respectively.

The following groups will be used for treatment period 1:

- AIN457 300 mg (2mL PFS): all subjects who are randomized to 300 mg 2mL PFS group at Randomization visit
- AIN457 300 mg (2x1mL PFS): all subjects who are randomized to 300 mg 2x1mL PFS group at Randomization visit
- Placebo: all subjects who are randomized placebo group at Randomization visit
- Any AIN457 300 mg: Any AIN457 300 mg of (2mL PFS) or (2x1mL PFS) as above.

The following groups will be used for entire treatment period:

- AIN457 300 mg (2mL PFS): all subjects who are randomized to 300 mg 2mL PFS group at Randomization visit
- AIN457 300 mg (2x1mL PFS): all subjects who are randomized to 300 mg 2x1mL PFS group at Randomization visit
- Any AIN457 300 mg (2mL PFS): all subjects who are randomized to 300 mg 2mL PFS group at Randomization visit and all placebo subjects who are re-assigned to 300 mg 2mL PFS at Week 12, but they are only considered after the treatment reassignment (Week 12 treatment injection).

- Any AIN457 300 mg (2x1mL PFS): all subjects who are randomized to 300 mg 2x1mL PFS group at Randomization visit and all placebo subjects who are re-assigned to 300 mg 2x1mL PFS at Week 12, but they are only considered after the treatment reassignment (Week 12 treatment injection).
- **Placebo**: all subjects who are re-assigned will only be considered until the reassignment point (Week 12 treatment injection).
- Any AIN457 300 mg: Any AIN457 300 mg of (2mL PFS) or (2x1mL PFS) as above.

## 2.8.1 Adverse events (AEs)

For adverse events and other binary safety variables crude incidence and exposure time-adjusted incidence will be derived as described below and summarized in Table 2-7.

All adverse events are summarized based on treatment emergent only. The definition for "treatment emergent" is as below:

- events started after the first dose of study medication or events present prior to the first dose of study medication but increased in severity based on preferred term
- and started prior to the last dose plus 84 days (inclusive)

All adverse events will be listed with "treatment emergent" flag displayed.

Table 2-7 Overview of analyses on some safety endpoints

| Analysis period | AEs &<br>SPP/RMP<br>risks<br>(special AE<br>interest) | SAEs | AEs-SMQ | AEs by<br>severity | study treatment<br>related AEs,<br>death & other<br>significant AEs | notables<br>(lab/vitals) |
|---|---|---|---|---|---|---|
| treatment<br>period 1<br>(up to<br>week 12) | •crude<br>incidence | •crude incidence | •crude incidence | •crude incidence | •crude<br>incidence | •crude incidence |
| Entire treatment<br>period<br>(including all<br>data) | <ul><li>crude<br/>incidence</li><li>exp.time<br/>adjusted<br/>incidence*</li></ul> | <ul> <li>crude<br/>incidence</li> <li>exp.time<br/>adjusted<br/>incidence*</li> </ul> | <ul><li>crude<br/>incidence</li><li>exp.time<br/>adjusted<br/>incidence*</li></ul> | • crude incidence | • crude<br>incidence | • crude incidence |

<sup>\*</sup>Note, Exposure adjusted incidence rates will be provided and follow the guideline as below:

- Primary SOC level for AE and SAE
- Level 1 for risks and SMQ
- PT level for SAE
- PT level for AE  $\geq$  2% or incidence rate per 100 subject years  $\geq$  5.0 in any treatment group
- Other selected AEs of special interest on lower levels (e.g. PT or SMQ level 2), if appropriate

The crude incidence of treatment emergent adverse events will be presented for the treatment period including all data

for final analysis. The crude incidence of treatment emergent adverse events will be summarized by primary System Organ Class (SOC) and Preferred Term (PT). Confidence intervals for the crude rate will be derived using the score method including continuity correction (Newcombe 1998) as described in Section 5.4.5. In addition, exposure time-adjusted incidence rates will be provided for the treatment period including all data (see Section 5.4.6).

Adverse events will be summarized by presenting, for each treatment group, the number and percentage of subjects having at least one AE, having an AE in each primary system organ class and having each individual AE (preferred term). Summaries will also be presented for AEs by severity and for study treatment related AEs. If a particular AE 'severity' is missing, this variable will be listed as missing and treated as missing in summaries. If a subject reported more than one adverse event with the same preferred term, the adverse event with the greatest severity will be presented. If a subject reported more than one adverse event within the same primary system organ class, the subject will be counted only once with the greatest severity at the system organ class level, where applicable.

Adverse events will also be summarized by standardized or customized MEdDRA queries (SMQ or CMQ/NMQ). The MedDRA version used for reporting the adverse events will be described in a footnote.

The most common adverse events reported ( $\ge z$  % in any group for each preferred term in the table by SOC and PT or  $\ge z$  % in any group for each grouping term table) will be presented in descending frequency according to its incidence in secukinumab group starting from the most common event. Here threshold value z is set to 2 (%) but it may be updated following review of the dry run outputs.

A graphical display of the crude rates or exposure adjusted incidence rates within system organ classes will be presented as follows: For all AEs regardless of severity and seriousness, the point estimate within system organ classes will be presented graphically with system organ class on the y-axis. This figure will consist of two panels: i) point estimate of AEs, ii) point estimate of serious AEs. For the exposure adjusted incidences a linear-scale will be used on the x-axes.

Separate summaries will be provided for deaths, serious adverse events, other significant adverse events leading to discontinuation and adverse events leading to dose adjustment or interruption.

Algorithms for date imputations will be provided in Section 5.

For SAEs occurred during screening a listing will be prepared for all subjects screened including screening failures.

The adverse events occurred after the treatment errors in those subjects who received erroneously the wrong treatment at least once, will be listed.

Other safety topics of interest, such as risks defined in the Safety Profiling Plan, Risk Management Plan or topics of interest regarding signal detection or routine analysis are defined

#### in the Program Case Retrieval Sheet

Crude rate of important identified and potential risks from Case Retrieval Sheet will be provided for all (non-serious and serious) cases and for all serious cases. Exposure-time adjusted rates will be provided for treatment period including all data for all (non-serious and serious) cases and for all serious cases. In addition, listings will be provided for the related AE risks.

Risk measures and confidence intervals will be derived according to Section 5.

The version of the Case Retrieval Sheet used for the analyses will be described in a footnote. This includes MedDRA version and Novartis MedDRA Query (NMQ) dictionary date.

**Important note:** For the evaluation of risks primary and secondary system organ classes of the MedDRA dictionary will be considered.

For the legal requirements of ClinicalTrials.gov and EudraCT, two required tables on adverse events which are not serious adverse events with an incidence greater than 2% and on serious adverse events and SAE suspected to be related to study treatment will be provided by system organ class and preferred term on the safety set population.

If for a same patient, several consecutive AEs (irrespective of study treatment causality, seriousness and severity) occurred with the same SOC and PT:

- a single occurrence will be counted if there is  $\leq 1$  day gap between the end date of the preceding AE and the start date of the consecutive AE
- more than one occurrence will be counted if there is > 1 day gap between the end date of the preceding AE and the start date of the consecutive AE

For occurrence, the presence of at least one SAE / SAE suspected to be related to study treatment / non SAE has to be checked in a block e.g., among AE's in a  $\leq$  1 day gap block, if at least one SAE is occurring, then one occurrence is calculated for that SAE.

The number of deaths resulting from SAEs suspected to be related to study treatment and SAEs irrespective of study treatment relationship will be provided by SOC and PT.

## 2.8.2 Deaths

Separate summary and listing will be provided for deaths.

## 2.8.3 Laboratory data

The summary of laboratory evaluations will be presented for two groups of laboratory tests (hematology and serum chemistry).

Descriptive summary statistics for the change from baseline to each study visit will be presented by laboratory test and treatment group. Change from baseline will only be summarized for subjects with both baseline and post baseline values and will be calculated as:

change from baseline = post baseline value – baseline value

Only "on-treatment" laboratory data will be summarized (i.e. assessments within last dose plus 84 days). All laboratory data will be listed with "on-treatment" flag displayed. If two

measurements are taken on the same date/time/CRF visit then use the average of two assessments.

For laboratory test values below Lower Level of Quantification (LLQ) or above Upper Level of Quantification (ULQ) will be imputed as LLQ or ULQ value, respectively. The numerical part of the reported result will be treated as the actual LLQ or ULQ. These laboratory values will be displayed in listings using the standard unit with the reported sign ("<" or ">")." For example, the actual lab result is "<5" and LLQ = 10, it will be reported for the numerical part as 5 and listed as "<5", LLQ will be imputed as 5.

In addition, shift tables may be provided as required at ad-hoc basis for all parameters to compare a subject's baseline laboratory evaluation relative to the most extreme laboratory test value within a treatment period. For the shift tables, the normal laboratory ranges will be used to evaluate whether a particular laboratory test value is normal, low, or high (including category "high and low"). These summaries will be presented by laboratory test and treatment group. Subjects with abnormal laboratory values will be listed and values outside the normal ranges will be flagged.

The following laboratory parameters will be analyzed with respect to numerical Common Terminology Criteria for Adverse Events (CTCAE) grades, given in Table 2-8: hemoglobin, platelets, white blood cell count, neutrophils, lymphocytes, creatinine, total bilirubin (TBL), gamma-glutamyl transferase (GGT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP).

The number and percentage of subjects with CTCAE grade newly occurring or worsening after baseline will be presented. These summaries will be split into hematology and chemistry.

Table 2-8 CTCAE grades for laboratory parameters to be analyzed

| CTCAE v4.0 Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| HGB decreased<br>(Anemia) | <lln 100="" g="" l<="" td="" –=""><td>&lt;100 – 80 g/L</td><td>&lt;80 g/L</td><td>Life-threatening consequences; urgent intervention</td></lln> | <100 – 80 g/L | <80 g/L | Life-threatening consequences; urgent intervention |
| Platelet count decreased | <lln 75.0="" l<="" td="" x10e9="" –=""><td>&lt;75.0 - 50.0 x10e9 /L</td><td>&lt;50.0 – 25.0 x10e9 /L</td><td>&lt;25.0 x 10e9 /L</td></lln> | <75.0 - 50.0 x10e9 /L | <50.0 – 25.0 x10e9 /L | <25.0 x 10e9 /L |
| White blood cell decreased | <lln -="" 10e9="" 3.0="" l<="" td="" x=""><td>&lt;3.0 - 2.0 x 10e9 /L</td><td>&lt;2.0 - 1.0 x 10e9 /L</td><td>&lt;1.0 x 10e9 /L</td></lln> | <3.0 - 2.0 x 10e9 /L | <2.0 - 1.0 x 10e9 /L | <1.0 x 10e9 /L |
| Neutrophil count decreased | <lln -="" 1.5="" 10e9="" l<="" td="" x=""><td>&lt;1.5 - 1.0 x 10e9 /L</td><td>&lt;1.0 - 0.5 x 10e9 /L</td><td>&lt;0.5 x 10e9 /L</td></lln> | <1.5 - 1.0 x 10e9 /L | <1.0 - 0.5 x 10e9 /L | <0.5 x 10e9 /L |
| Lymphocyte count decreased | <lln -="" 0.8="" 10e9="" l<="" td="" x=""><td>&lt;0.8 - 0.5 x 10e9 /L</td><td>&lt;0.5 - 0.2 x 10e9 /L</td><td>&lt;0.2 x 10e9 /L</td></lln> | <0.8 - 0.5 x 10e9 /L | <0.5 - 0.2 x 10e9 /L | <0.2 x 10e9 /L |
| Creatinine increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 6.0 x ULN | >6.0 x ULN |
| TBL increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| ALT increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| AST increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| ALP increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |

Shift tables will be presented comparing baseline laboratory result (CTCAE grade) with the worst results (expressed in CTCAE grade) during the treatment phase analyzed. Of note, baseline will be defined as last assessment prior to first dosing in initial treatment phase. If no

pre-treatment value exists, also a value recorded after first dose can be used as baseline if it was collected on the same day as first dose, see Section 2.1.1.3.

Exposure time adjusted incidence for subjects with newly occurring neutropenia of CTCAE grade >=2 will be summarized and listed in the listing.

The number and percentage of subjects with newly occurring liver enzyme abnormalities will also be summarized based on the event criteria given in Table 2-9.

Table 2-9 Liver-related events

| Table 2-9 | Liver-related events |
|---|---|
| Parameter | Criterion |
| ALT | >3xULN; >5xULN; >8xULN;>10xULN, >20xULN |
| AST | >3xULN; >5xULN; >8xULN; >10xULN; >20xULN |
| ALT or AST | >3xULN; >5xULN; >8xULN; >10xULN; >20xULN |
| | ALT or AST >3xULN & (nausea or vomiting or fatigue or general malaise or abdominal pain or (rash and eosinophilia)) |
| TBL | >1xULN;>1.5xULN; >2xULN; >3xULN, |
| ALP | >1.5xULN;>2xULN; >3xULN; >5xULN |
| ALT or AST & | ALT or AST>3xULN & TBL >1.5xULN; |
| TBL | ALT or AST>3xULN & TBL >2xULN; |
| | ALT or AST >5xULN & TBL >2xULN; |
| | ALT or AST >8xULN & TBL >2xULN; |
| | ALT or AST >10xULN & TBL >2xULN; |
| | ALT or AST >20xULN & TBL >2xULN; |
| ALP & TBL | ALP >3xULN & TBL >2xULN |
| | ALP >5xULN & TBL >2xULN |
| ALT or AST & | ALT or AST>3xULN & TBL >2xULN & ALP <2xULN (Potential Hy's Law) |
| TBL & ALP | Note: elevated ALP may suggest obstruction as a consequence of gall bladder or bile duct disease; ALP may also be increased in malignancy. FDA therefore terms Hy's Law cases as indicators of <i>pure hepatocellular injury</i> . This does not mean that cases of ALT or AST >3xULN & TBL >2xULN & ALP ≥2xULN may not result in severe DILI. |
| | ALT or AST>3xULN & TBL >2xULN & ALP <2xULN ( <b>Potential Hy's Law</b> ) or reported Hy's Law case |
| | Note: "Hy's Law case" is a lower level term in MedDRA (10070546) and may be reported as AE. |

For a combined criterion to be fulfilled, all conditions have to be fulfilled on the same visit. The criteria are not mutually exclusive, e.g., a subject with ALT = 6.42xULN is counted for ALT > 3xULN and ALT > 5xULN.

Individual subject data listings will be provided for subjects with newly occurring or worsening abnormal laboratory data. Data of subjects with newly occurring liver enzyme abnormalities will be listed in an additional listing.

Fasting laboratory tests including fasting plasma glucose and fasting lipids will be evaluated only at screening. No analysis will be done for these measurements.

For urinalysis, standard dipstick measurements for specific gravity, protein, glucose, pH, blood, urine blood (non-hemolyzed), urine blood (hemolyzed), bilirubin, ketones, WBC will be done at screening. No analysis will be done for these measurements.

#### 2.8.4 Other safety data

## 2.8.4.1 ECG and cardiac imaging data

A standard 12-lead ECG will be performed at screening to assess the eligibility of subjects. No analysis will be done for ECG measurements.

#### 2.8.4.2 Vital signs

Analysis in vital sign measurement using descriptive summary statistics for the change from baseline for each post-baseline visit will be performed by vital sign and treatment group. Change from baseline will only be summarized for subjects with both baseline and post-baseline values and will be calculated as:

change from baseline = post-baseline value – baseline value

Only "on-treatment" vital signs will be summarized (i.e. assessments within last dose plus 84 days). All vital signs will be listed with "on-treatment" flag displayed.

The number and percentage of subjects with newly occurring notable vital signs abnormalities will be presented. Criteria for notable vital sign abnormalities are provided in Table 2-10 below. A listing of subjects with newly occurring notably abnormal vital signs will be provided.

Table 2-10 Criteria for notable vital sign abnormalities

| Vital sign (unit) | Notable abnormalities |
|---------------------------------|--------------------------|
| Systolic blood pressure (mmHg) | >= 140 mmHg or < 90 mmHg |
| Diastolic blood pressure (mmHg) | >=90 mmHg or <60 mmHg |
| Pulse (bpm) | > 100 bpm or <60 bpm |

#### 2.9 Pharmacokinetics

All completed subjects with quantifiable secukinumab serum concentration will be included in the pharmacokinetic data analysis.

Serum concentrations will be expressed in mass per volume units. All concentrations below the limit of quantification as well as missing data will be labeled as such in the concentration data listings.

Secukinumab serum concentrations will be summarized by visit and treatment group. In addition to mean, standard deviation (SD), coefficient of variation (CV), median and quartiles, the geometric mean and geometric coefficient of variation (CV) and n(log) will be presented. The formula for deriving the geometric mean and CV (%) is as following:

- CV (%) = (SD/mean)\*100,
- geometric mean=exp( (sum of log transformed data) / number of non-missing data points after log transformation),
- geometric CV = sqrt( exp( variance of log-transformed data)-1)\*100.

Secukinumab serum concentration in the AIN457 300mg (2mL PFS) group will also be summarized by injections locations at previous 3 visits (i.e., though only, abdomen only, and though and abdomen) at Weeks 28 and 52. For Week 28, the previous injections locations at Weeks 16, 20 and 24 will be considered. Likewise for Week 52, the previous injections locations will be at Weeks 40, 44 and 48.

In addition, concentration, sample date, sample time at pre-dose and minutes pre-dose, elapse time since day of first secukinumab dose, reason excluding from analysis will be listed by treatment sequence. Placebo subjects will also be listed.

Values below lower limit of quantification/below detection limit will be imputed by 0.

The analysis visit will refer to the visit as per the CRF.

Pharmacokinetic parameters will be summarized by treatment group (AIN457 300mg 2mL PFS and AIN457 300 mg 2×1mL PFS). Descriptive summary statistics for Cmax and AUC84-112d include mean (arithmetic and geometric), SD, and CV (arithmetic and geometric), median, minimum and maximum. Tmax in days will be summarized as median, minimum and maximum. In addition, pharmacokinetic parameters will be listed by treatment sequence.

The log-transformed parameters Cmax and AUC84-112d will be analyzed by a linear model, with treatment group (AIN457 300mg 2mL PFS and AIN457 300 mg 2×1mL PFS) as a fixed factor and body weight at baseline as covariate. For each of Cmax and AUC84-112d, the mean estimate and 90% confidence interval for the PK parameter ratio of "AIN457 300mg 2mL PFS" vs "AIN457 300 mg 2×1mL PFS" will be reported to represent the relative bioavailability for comparison. The log-transformed AUC84-112d at Week 12 in the AIN457 300mg (2mL PFS) group will be analyzed by a linear model, with injection location, laterality and body weight at baseline. The mean estimate and 90% confidence interval for the ratio of thigh vs abdomen and that of left vs right will be reported.

In addition, a linear model with previous injections locations and body weight at baseline will be fitted for the log-transformed AUC84-112d at Week 12 in the AIN457 300mg (2mL PFS) group. The mean estimate and 90% confidence interval for the ratio of "thigh only" vs "abdomen only", and that of "thigh and abdomen" vs "abdomen only" will be reported. For Week 12, the previous injections locations at randomization, Weeks 1, 2, 3, 4 and 8 will be considered.

## 2.11 Clinician-reported outcomes

#### 2.11.1 Usability and hazard assessment of the 2 mL pre-filled syringe

This analysis will be based on the Safety Set.

The number and percentage of subjects who successfully completed each and ALL of the indicated steps as per the IFU will be summarized by visit and treatment group, including total.

The number and percentage of subjects who experienced each and ANY of the defined possible hazards will be summarized by visit and treatment group, including total.

Successful self-injection will be positively defined for a subject when the subject performs the six critical steps as per the IFU (i.e. P8, P10, P11, P12, P13, P14). Number and percentage of subjects who passed the self-injection successfully as well as a two-sided 95% exact confidence interval at Week 1 visit will be summarized by visit and treatment group, including total. The following statistical hypothesis will be tested by an exact binomial test at one-sided 2.5% level of significance at Week 1 visit:

H<sub>0</sub>: successful pre-filled syringe use rate < 90%

 $H_1$ : successful pre-filled syringe use rate  $\geq 90\%$ 

Missing values with respect to the self-assessment checklist and possible hazard assessment checklist will not be imputed while summarizing the answers of each question with frequencies.

Subjects with one or more of the critical steps missing will be considered as unsuccessful (imputation with non-response) with regard to the self-injection success. Subjects who discontinued or who missed a visit and have the full self-injection checklist missing will not be evaluated with regard to the self-injection success at the corresponding visit.

Visit windows will not be applied to self-injection assessment and possible hazard assessment. The analysis visit will refer to the visit as per the CRF.

Of note: only data in the self-assessment checklist with self-injection checked in eCRF Dosage Administration Record (DAR) page are included in the analyses.

## 2.12 Patient-reported outcomes

Summaries will be based on the FAS and will be presented separately for each treatment group.

For DLQI missing values will be replaced by LOCF. Baseline values will not be carried forward. If no pre-treatment value exists, values obtained after first dose of treatment can be used as baseline only if it was collected on the same day as first dose. In addition, missing baseline (PROs) values will be replaced by the means or modes of non-missing baseline values stratified by age group (<65 years, 65 years and older) and sex, for continuous scale or categorical/ordinal scale, respectively.

### **Dermatology Life Quality Index**

The DLQI measures functional disability of subjects with dermatological disorders that are greater than 18 years of age and had been utilized as a relevant clinical measure in atopic dermatitis, as well as other dermatitis clinical trials. The DLQI is a simple, validated, self-administered 10-item questionnaire. The instrument contains six functional scales (i.e., symptoms and feeling, daily activities, leisure, work and school, personal relationships, treatment). For the DLQI, each question will be answered with the following response: "not at all", "a little", "a lot", or "very much". "Not relevant" is also a valid response. Seven scores will be derived from the DLQI: the total score of each of the six dimensions as well as the total score over all items. The higher the score, the more quality of life is impaired.

For each of the seven scores, the percentage change from baseline will be derived. Summary statistics will be provided for absolute values as well as for the percentage change by visit and treatment group.

In addition, summary statistics will be provided for number of subjects achieving DLQI 0 or 1. Treatment groups will be compared by Fisher's exact test.



## **Self-Injection Assessment Questionnaire (SIAQ)**

All SIAQ analyses will be based on the Safety Set.

Summary statistics for the absolute values of the domain scores at Randomization (baseline) will be provided by treatment group including total for the PRE-module and the POST-module. The number and percentage of subjects in each of the 5 categories (likert scale) for each item will be presented by visit and treatment group including total.

Item and domain scores from the PRE module taken before the first self-injection at Randomization (baseline) will be compared with the corresponding item and domain scores (feeling about injections, self-confidence domains, and overall satisfaction of self-injection item) from the POST modules. Change in domain scores from PRE module will be summarized by visit and treatment group including total.

Domain scores will be calculated only if 50% or more items of the domain are completed. Missing items will not be imputed. Subjects who discontinued or who missed a visit and have the SIAQ questionnaire not completed will not be considered in the analyses at the corresponding visit.

Of note: only SIAQ scores for those with self-injection checked in eCRF DAR page are included in the analyses.





## 3 Sample size calculation

A response rate of 8% for PASI 75 response and IGA mod 2011 0 or 1 response in the placebo group is expected, whereas a response rate of 62% for PASI 75 response and 55% for IGA mod 2011 0 or 1 is the anticipated response in the secukinumab 300 mg 2 mL pre-filled syringe group.

Placebo-response rates between 3% and 7% have been reported in Papp et al 2005, Menter et al 2008, Leonardi et al 2008, and Papp et al 2008.
# 3.1 Primary endpoint (co-primary endpoint)

With respect to the co-primary endpoint (PASI 75 response and IGA mod 2011 0 or 1 response at Week 12), the type-I-error will be 2.5% one-sided for comparison. With 70 subjects per group and assuming a response rate of 10% for PASI 75 response and IGA mod 2011 0 or 1 response in the placebo group, the power to show a response rate of 62% for PASI 75 response and 55% for IGA mod 2011 0 or 1 response in the secukinumab 300 mg 2 mL pre-filled group based on Fisher's exact test (nQuery Advisor 6.01, two group Fisher's-exact test of equal proportions) is above 99% for PASI 75 response and IGA mod 2011 0 or 1 response.

# 3.1.1 Secondary endpoints

A power of 90% to show a response rate of 30% for PASI 100 in the secukinumab 300 mg 2 mL pre-filled group and 8% in the placebo group based on Fisher's exact test results in a sample size of 70 subjects per group. Same power can be achieved if we apply the same assumption of PASI 100 response rate for secukinumab 300 mg 1 mL pre-filled group.

A power of above 99% to show a response rate of 46% for PASI 90 in the secukinumab 300 mg 2 mL pre-filled group and 8% in the placebo group based on Fisher's exact test results in a sample size of 70 subjects per group.

# 4 Change to protocol specified analyses

The primary and secondary efficacy endpoints will be analyzed using logistic regression model. Exact logistic regression will be performed in case of low response rates in the placebo group.

The following analyses have been removed:

- The maximum change (maximum decrease and maximum increase) from baseline within treatment period for each laboratory parameter
- The stratified Van-Eltern testing and Hodges-Lehmann estimates for the absolute value and the percentage change from baseline of DLQI total score.

# 5 Appendix

#### 5.1 Imputation rules

#### 5.1.1 Study drug

Any partial dates will be imputed as follows:

We take the earlier day of

- The last day in the month and
- The calculated end day of the corresponding epoch

#### 5.1.2 AE date imputation

#### Impute AE end date:

- 1. If the AE end date 'month' is missing, the imputed end date should be set to the earliest of the (min (last visit date, last dose date + 84 days), 31DECYYYY, date of death).
- 2. If the AE end date 'day' is missing, the imputed end date should be set to the earliest of the (min (last visit date, last dose date + 84 days), last day of the month, date of death).
- 3. If AE 'year' is missing or AE is ongoing, the end date will not be imputed.

### Impute AE start date:

Before imputing AE start date, find the AE start reference date.

- 1. If the (imputed) AE end date is complete and the (imputed) AE end date < treatment start date then AE start reference date = min(informed consent date, earliest visit date).
- 2. Else AE start reference date = treatment start date
- 1. If the AE start date 'year' value is missing, the date uncertainty is too high to impute a rational date. Therefore, if the AE year value is missing, the imputed AE start date is set to NULL.
- 2. If the AE start date 'year' value is less than the treatment start date year value, the AE started before treatment. Therefore:
  - a. If AE 'month' is missing, the imputed AE start date is set to the mid-year point (01JulYYYY).
  - b. Else if AE 'month' is not missing, the imputed AE start date is set to the mid-month point (15MONYYYY).
- 3. If the AE start date year value is greater than the treatment start date year value, the AE started after treatment. Therefore:
  - a. If the AE month is missing, the imputed AE start date is set to the year start point (01JanYYYY).

- b. Else if the AE month is not missing, the imputed AE start date is set to the later of (month start point (01MONYYYY), AE start reference date + 1 day).
- 4. If the AE start date year value is equal to the treatment start date year value:
  - a. And the AE month is missing the imputed AE start date is set to the AE reference start date + 1 day.
  - b. Else if the AE month is less than the treatment start month, the imputed AE start date is set to the mid-month point (15MONYYYY).
  - c. Else if the AE month is equal to the treatment start date month or greater than the treatment start date month, the imputed AE start date is set to the later of (month start point (01MONYYYY), AE start reference date + 1 day).

If complete (imputed) AE end date is available and the imputed AE start date is greater than the (imputed) AE end date, then imputed AE start date should be set to the (imputed) AE end date.

# 5.1.3 Concomitant medication date imputation

Impute CM end date:

- 1. If CM end day is missing and CM month/year are non-missing then impute CM day as the minimum of treatment end date and the last day of the month.
- 2. If CM end day/month are missing and CM year is non-missing then impute CM day as the minimum of treatment end date and the end of the year (31DECYYYY).
- 3. If imputed CM end date is less than the CM start date, use the CM start date as the imputed CM end date.

Impute CM start date:

- 1. If the CM start date year value is missing, the imputed CM start date is set to one day prior to treatment start date.
- 2. If the CM start date year value is less than the treatment start date year value, the CM started before treatment. Therefore:
  - a. If the CM month is missing, the imputed CM start date is set to the mid-year point (01JulYYYY).
  - b. Else if the CM month is not missing, the imputed CM start date is set to the midmonth point (15MONYYYY).

- 3. If the CM start date year value is greater than the treatment start date year value, the CM started after treatment. Therefore:
  - a. If the CM month is missing, the imputed CM start date is set to the year start point (01JanYYYY).
  - b. Else if the CM month is not missing, the imputed CM start date is set to the month start point (01MONYYYY).
- 4. If the CM start date year value is equal to the treatment start date year value:
  - a. And the CM month is missing or the CM month is equal to the treatment start date month, then the imputed CM start date is set to one day prior treatment start date.
  - b. Else if the CM month is less than the treatment start date month, the imputed CM start date is set to the mid-month point (15MONYYYY).
  - c. Else if the CM month is greater than the treatment start date month, the imputed CM start date is set to the month start point (01MONYYYY).

If complete (imputed) CM end date is available and the imputed CM start date is greater than the (imputed) CM end date, then imputed CM start date should be set to the (imputed) CM end date.

# 5.1.3.1 Prior therapies date imputation

See Section 5.1.3.

## 5.1.3.2 Post therapies date imputation

See Section 5.1.3.

#### 5.1.4 First diagnosis date (PsO, PsA) imputation

- 1. If the first diagnosis day/ month are missing and the year is non-missing:
  - a. If the year part of the first diagnosis date is equal to the year part of the inform consent date, then the imputed first diagnosis date is set to the year start point (01JanYYYY).
  - b. Otherwise the imputed first diagnosis date is set to the mid-year point (01JulYYYY).
- 2. If the first diagnosis day is missing and the month/year are non-missing:

a. If the month and year part of the first diagnosis date is equal to the month and year part of the inform consent date, then the imputed first diagnosis date is set to the month start point (01MONYYYY).

b. Otherwise the imputed first diagnosis date is set to the mid-month point (15MONYYYY).

# 5.1.5 Other imputations

Only PASI and IGA mod 2011 based response variables are imputed with multiple imputation or non-response, other response variables (e.g. DLQI 0 or 1 achievement) will be imputed with LOCF.

For DLQI, missing values will be replaced by LOCF. Baseline values will not be carried forward. If no pre-treatment value exists, values obtained after first dose of treatment can be used as baseline only if it was collected on the same day as first dose. In addition, missing baseline (PROs) values will be replaced by the means or modes of non-missing baseline values stratified by age group (<65 years, 65 years and older) and sex, for continuous scale or categorical/ordinal scale, respectively.

For laboratory test values below Lower Level of Quantification (LLQ) or above Upper Level of Quantification (ULQ) will be imputed as LLQ or ULQ value, respectively. The numerical part of the reported result will be treated as the actual LLQ or ULQ. These laboratory values will be displayed in listings using the standard unit with the reported sign ("<" or ">")."

# 5.2 AEs coding/grading

Adverse events will also be coded according to MedDRA dictionary, using a narrow search. The MedDRA version used for reporting the adverse events will be described in a footnote.

Safety topics of interest, such as risks defined in the Safety Profiling Plan, Risk Management Plan or topics of interest regarding signal detection or routine analysis are defined in the Program Case Retrieval Sheet

# 5.3 Laboratory parameters derivations

See Section 2.8.3.

#### 5.4 Statistical models

#### 5.4.1 Analysis of continuous data

Summary statistics (including N, mean, standard deviation, minimum, lower quartile, median, upper quartile, maximum) will be provided for continuous data by visit and treatment group. For PASI score, DLQI total scores, summary statistics will be derived for absolute and percentage changes from baseline.

# 5.4.2 Analysis of binary (and categorical) data

Summary statistics for discrete variables will be presented in contingency tables and will include absolute and relative frequencies. If applicable, confidence intervals will be derived as well based on the score method including continuity correction [Newcombe (1998)]:

With z as (1-alpha/2)-quantile of the standard normal distribution (SAS: z=PROBIT(1-alpha/2), n as total number of subjects (i.e. number of subjects in the denominator), and p as estimated crude incidence (number of subjects with event n) it is q = 1 - p

Then the lower limit is for p > 0, (L = 0 for p = 0),

$$L = \max\left(0, \frac{2np + z^2 - 1 - z\sqrt{z^2 - 2 - \frac{1}{n} + 4p(nq + 1)}}{2(n + z^2)}\right)$$

and the upper limit is for p < 1, (U = 1 for p = 1),

$$U = \min \left(1, \frac{2np + z^2 + 1 + z\sqrt{z^2 + 2 - \frac{1}{n} + 4p(nq - 1)}}{2(n + z^2)}\right).$$

For response variables (e.g. for IGA mod 2011 0 or 1, PASI 75, PASI 50, PASI 90 and PASI 100 response) the placebo adjusted response rates (risk difference) including 95% confidence interval will be derived by visit.

Figures will be provided for PASI 75 response (upper left) PASI 90 response (upper right), PASI 100 response (lower left) and IGA mod 2011 0 or 1 response (lower right) at Week 12 as dot plots displaying treatments on the x-axis and point estimates including 95% confidence intervals on the y-axis.

For time courses of response variables, the point estimate at each time point including 95% confidence interval will be plotted.

# 5.4.3 Logistic regression

Binary outcome variables, including PASI 50 / 75 / 90 / 100 response and IGA mod 2011 0 or 1 response, will be evaluated using a logistic regression model with treatment regimen, baseline bodyweight and baseline PASI score. Odds ratios will be computed for comparisons of secukinumab dose regimen versus placebo utilizing the logistic regression model fitted.

If response rates are 0% or 100% in one of the treatment groups odds ratio estimate and p-values will not be displayed in outputs, but "-" will be shown.

The odds ratio will be calculated such that an odds ratio >1 is favorable for secukinumab. Using PROC GENMOD to calculate the confidence interval for the odds ratios assumes asymptotic normality of the Wald estimate for the regression coefficient. The 95% confidence interval for the regression parameter of the active treatment effect relative to control(s) will be calculated using an exponential transformation to create the confidence interval for the odds ratio.

All p-values reported on linear hypotheses about regression coefficients will be based on the Wald tests from Type III analyses. In the SAS procedure PROC GENMOD, a Type III analysis will be performed by adding the model options: TYPE3, DIST=BIN, and LINK=LOGIT.

Logistic regression will be applied to response variables at each visit.

If logistic regression model does not converge, the following steps will be performed:

- 1. Run the PROC GENMOD procedure with EXACT statement;
- 2. If convergence not reached, remove the covariates from the model one by one until convergence is reached; start with continuous covariates (i.e., baseline bodyweight by replacing with body weight stratum, and then baseline PASI score), followed by removing categorical covariates (i.e., weight stratum);
- 3. If convergence not reached, perform Fisher's exact test.

It should be noted that this model might not converge if response rates are too low.

#### 5.4.4 Multiple imputations for response variables

Primary and secondary endpoints will be evaluated by Logistic regression and odds ratio estimate as described in the primary analysis method with multiple imputations for missing values. In addition, logistic regression analysis for PASI 50, PASI 75, PASI 90, PASI 100 and IGA mod 2011 0 or 1 response by visits will be analyzed using multiple imputation method.

In the multiple imputations analysis the response status will be imputed based on the individual treatment arm information.

Multiple imputation (MI) is a simulation based approach where missing values are replaced by multiple Bayesian draws from the conditional distribution of missing data given the observed data and covariates, creating multiple completed data sets. These completed data sets can then be analyzed using standard methods. Rubin (1987) presented rules how to combine the multiple sets of estimates to produce overall estimates and confidence intervals that adequately incorporate missing data uncertainty.

Missing values for the 'change from baseline PASI score' and 'IGA mod 2011 score' will be imputed simultaneously based on an underlying joint normal distribution and using a Markov Chain Monte Carlo (MCMC) method. The change from baseline in PASI score appears to follow closer to a normal distribution than the actual PASI score. Assuming normality for the 'IGA mod 2011 score' is motivated by Schaefer (1997), where it was shown that the multivariate normal approximation for the imputation of incomplete categorical and binary data is robust.

The imputations will be done separately for each treatment group including baseline weight, failure to at least one previous biologic (yes/no), and number of previous systemic therapies as additional covariates.

Summary statistics for PASI 50, PASI 75, PASI 90, PASI 100, and IGA mod 2011 0 or 1 response by visit will be presented in contingency tables with multiple imputations method.

The number of imputations will be set to 100, the seed for the random function will be set to 4572323 for this study. To generate the multiple imputed data sets, the SAS procedure MI can be used as follows:

The input data set <pasi\_iga> should have one record per subject with baseline PASI score and IGA mod 2011 score as well as all changes from baseline PASI and post-baseline IGA mod 2011 score.

#### Programming notes:

- The SAS procedure MIANALYZE expects a variable called "\_IMPUTATION\_ which is generated by the MI procedure. It might be needed to set the SAS option "VALIDVARNAME=UPCASE" temporarily in the program before the MI call, this option should be reset after the MIANALYZE call to VALIDVARNAME=V6.
- In case there are no missings in one treatment group, the MI procedure does not impute any values. In this case the corresponding data need to be imputed manually outside PROC MI and added to the dataset <impdata>.

The imputed data are saved in data set <impdata>. The outcomes of interest, i.e. the PASI 50/75/90/100 response and IGA mod 2011 0 or 1 response will be calculated, e.g. as follows:

```
DATA <impdata2>;
SET <impdata>;
IF <change from baseline PASI week primary endpoint>/<baseline PASI>=0.75 THEN <PASI 75 response> =1;
ELSE <PASI 75 response>=0;
<...repeat for all PASI response...>
IF <baseline IGA> >=3 THEN DO;
         IF <IGA week primary endpoint> < 1.5 THEN <IGA 0/1 response> =1;
    ELSE IF <IGA week primary endpoint> >=1.5 THEN <IGA 0/1 response> =0;
    ELSE PUT "E" "RROR:" stysid1a=;
END:
ELSE IF <baseline IGA>=2 THEN DO;
         IF <IGA week primary endpoint> < 0.5 THEN <IGA 0/1 response> =1;
    ELSE IF <IGA week primary endpoint> >=0.5 THEN <IGA 0/1 response> =0;
    ELSE PUT "E" "RROR:" stysid1a=;
ELSE <IGA 0/1 response> =0;
RUN;
```

The treatment differences for each imputed data set will then be evaluated by Logistic regression and ODDS ratio as described in Section 5.4.6.2. This analysis will be done by

\_IMPUTATION\_ for the comparison to the placebo treatment group. The model should be estimating response probability = 1 by using DESECENDING option. Using the ESTIMATE option in the GENMOD procedure and the ODS OUTPUT data set "Estimates" provides the estimate for the odds ratio and confidence intervals.

```
PROC GENMOD <option>;
CLASS <stratum> <treatment>;
MODEL <response> = <explanatory variables> / link=logit dist=bin type3;
BY <by-variables);
ESTIMATE "OR. AIN 300 mg 2mL PFS VS. Placebo" <treatment> 1 0 -1/exp;
ESTIMATE "OR. AIN 300 mg 2x1mL PFS VS. Placebo" <treatment> 0 1 -1/exp;
ODS OUTPUT Estimates=Estimates;
RUN:
```

The MIANALYZE procedure expects the parameter estimate in the variables ESTIMATE, and the corresponding standard error in the variable STDERR. Measurements can be obtained from "Estimates" dataset by selecting the row with ODDS ratio estimates.

```
Data <modified dataset>;
  set Estimates;
  if substr(label,1,3)= "Exp";
  ESTIMATE=LBetaEstimate;
  STDERR=StdErr;
  effect= "OR";
  if missing(ESTIMATE) or missing(STDERR) then delete;
RUN:
```

The estimates and standard errors based on the 100 imputed data are then combined by applying Rubin's rules for multiple imputed data sets, see Little and Rubin (2002).

#### Programming notes:

- The variables ESTIMATE and STDERR in the input data set for the MIANALYZE procedure may not be missing. Records with missing values need to be deleted and the variable \_IMPUTATION\_ needs to be renumbered and regenerated since for each bygroup the procedure expects consecutive numbers starting at 1.
- The ESTIMATE and STDERR in terms of odds ratios from logistic regressions will be transformed to follow a normal distribution before MIANALYZE procedure. They will be transformed back to Odds Ratio to get the corrected ESTIMATE and corresponding CIs.

The SAS procedure MIANALYZE will be applied as follows:

```
DATA <modified dataset_t>;
    SET <modified dataset>;
    estimate=log(ESTIMATE);
    stderr=(log(LBETAUPPERCL)-log(LBETALOWERCL))/(2*1.96);
RUN;

ODS LISTING CLOSE;
ODS OUTPUT ParameterEstimates=<results> VarianceInfo=<varinfo> ModelInfo=<modelinfo>;
PROC MIANALYZE PARMS=<modified dataset>;
    BY <by-variables>;
    MODELEFFECTS ESTIMATE;
```

```
SETDERR stderr;
RUN;
ODS LISTING;

data <results_back>;
    set <results>;
    estimate=exp(ESTIMATE);
    LCLMEAN=estimate*exp(-1.96*stderr);
    UCLMEAN=estimate*exp(+1.96*stderr);
RUN;
```

In case if logistic regression does not converge, risk difference estimates will be provided. The SAS procedure PROC FREQ for risk difference estimates will be applied as follows:

```
ODS LISTING CLOSE;
PROC FREQ DATA=<Imputed dataset> ORDER=DATA;
     TABLES <treatment group>*<response variable>/riskdiff alpha=0.05;
     BY <By-variables>;
     ODS OUTPUT RiskDiffCol1=RiskDiffCol1;
RUN;
ODS LISTING;
DATA DRISK; SET RiskDiffCol1;
     WHERE control= "1";
     ESTIMATE=risk;
     STDERR=ase;
     effect="Riskdiff";
     IF missing(ESTIMATE) OR missing(STDERR) THEN DELETE;
RUN;
PROC SORT DATA=DRISK; BY <By-variables>; RUN;
ODS LISTING CLOSE;
ODS OUTPUT ParameterEstimates=results VarianceInfo=varinfo ModelInfo=Modelinfo;
PROC MIANALYZE PARAMS=drisk;
    by <By-variables>;
     modeleffects Riskdiff;
     stderr ase;
RUN;
ODS LISTING;
DATA results2;
    set results;
     or=estimate*100;
     lowercl=(LCLmean)*100;
     uppercl=(UCLmean)*100;
     KEEP <response variable> <By-variables> or lowercl uppercl probt;
RUN;
```

### 5.4.5 Crude incidence and related risk estimates

### 5.4.5.1 Crude incidence and 100\*(1-α)% confidence interval

For n subjects, each at risk to experience a certain event with probability  $\pi$ , the crude incidence is estimated as p=x/n, where x is the number of subjects with the event.

Absolute and relative frequencies will be displayed as well as 95% confidence interval for the relative frequency based on the score method including continuity correction (Newcombe 1998).

With z as  $(1-\alpha/2)$ -quantile of the standard normal distribution (SAS: z=PROBIT(1-alpha/2), n as total number of subjects (i.e. number of subjects in the denominator), and p as estimated crude incidence (number of subjects with event / n) it is q = 1 - p.

Then the lower limit is

$$L = \max\left(0, \frac{2np + z^2 - 1 - z\sqrt{z^2 - 2 - \frac{1}{n} + 4p(nq + 1)}}{2(n + z^2)}\right)$$

and the upper limit is

$$U = \min\left(1, \frac{2np + z^2 + 1 + z\sqrt{z^2 + 2 - \frac{1}{n} + 4p(nq - 1)}}{2(n + z^2)}\right).$$

Note: if p = 0 then L = 0 and if p = 1 then U = 1.

If appropriate, an exact  $100*(1-\alpha)\%$  confidence interval (Clopper-Pearson 1934) will be obtained by using the SAS procedure PROC FREQ with the EXACT BINOMIAL statement. However, the confidence interval derived via the score method including continuity correction will be the default in safety analyses.

## 5.4.5.2 Relative risk and 100\*(1-α)% confidence interval

For an investigational drug group with  $n_1$  subjects at risk, independent from the control group (e.g., placebo or comparator) with  $n_0$  subjects at risk, of whom  $x_1$  and  $x_0$  experience a certain event with probability  $\pi_1$  and  $\pi_0$  respectively, the relative risk is estimated as  $p_1/p_0$  with  $p_1=x_1/n_1$  and  $p_0=x_0/n_0$ .

An asymptotic  $100*(1-\alpha)\%$  confidence interval on the relative risk will be based on the backtransformed large sample confidence limits on the log-transformed relative risk estimate which are obtained by application of the delta-method and Slutzky's theorem (Lachin 2000). The SAS procedure PROC FREQ with option RELRISK in the TABLES statement will be used to provide the asymptotic  $100*(1-\alpha)\%$  confidence interval on the relative risk. The estimate is not computed if either  $x_1$  or  $x_0$  equals 0. In this case, or if the crude incidences are low in both groups, the relative risk will be approximated by the odds ratio for which an exact confidence interval will be obtained as specified in Section 5.4.6.3. If the relative risk is not well approximated by the odds ratio but asymptotic normality is questionable, STATXACT will be used.

#### 5.4.5.3 Odds ratio and 100\*(1-α)% confidence interval

For an investigational drug group with  $n_1$  subjects at risk, independent from the control group (e.g. placebo) with  $n_0$  subjects at risk, of whom  $x_1$  and  $x_0$  experience a certain event with probability  $\pi_1$  and  $\pi_0$  respectively, the odds ratio is estimated as

 $\frac{p_1/(1-p_1)}{p_0/(1-p_0)}$  with  $p_1=x_1/n_1$  and  $p_0=x_0/n_0$ . A conditional exact  $100*(1-\alpha)\%$  confidence interval

will be obtained by using the SAS procedure PROC FREQ with statement EXACT OR.

# 5.4.5.4 Risk difference and 100\*(1-α)% confidence interval

For an investigational drug group with  $n_1$  subjects at risk, independent from the control group (e.g., placebo or comparator) with  $n_0$  subjects at risk, of whom  $x_1$  and  $x_0$  experience a certain event, the risk difference is estimated as  $p_1$ - $p_0$  with  $p_1$ =  $x_1/n_1$  and  $p_0$ = $x_0/n_0$ .

Exact unconditional confidence limits for the risk difference will be obtained with SAS procedure PROC FREQ and option RISKDIFF in the TABLES statement, specifying the RISKDIFF option also in the EXACT statement.

### 5.4.6 Exposure adjusted incidence rate and related risk estimates

# 5.4.6.1 Exposure adjusted incidence rate and 100\*(1-α)% confidence interval

It will be assumed that for each of n subjects in a clinical trial the time  $t_j$  (j=1,...,n) to the first occurrence of a certain treatment emergent event is observed, or if the event was not experienced, the (censored) time to the end of the observation period or last dose plus 84 days whichever occur earlier. The sequence of first occurrences of an event will be modeled to follow approximately a Poisson process with constant intensity  $\theta$ . The rate parameter  $\theta$  will be

estimated as  $\lambda = D/T$ , where  $T = \sum_{j=1}^{n} t_j$  and D is the number of subjects with at least one event.

Conditionally on T, an exact  $100*(1-\alpha)\%$  confidence interval for a Poisson variable with parameter  $\theta T$  and observed value D can be obtained based on (Garwood, 1936), from which an exact  $100*(1-\alpha)\%$  confidence interval for D/T will be derived as follows (Sahai, 1993; Ulm, 1990):

Lower confidence limit  $L = \frac{0.5c_{\alpha/2,2D}}{T}$  for D>0, 0 otherwise,

Upper confidence limit 
$$U = \frac{0.5c_{1-\alpha/2,2D+2}}{T}$$

where  $c_{\alpha,k}$  is the  $\alpha$ th quantile of the Chi-square distribution with k degrees of freedom.

#### 5.4.6.2 Exposure-adjusted event rate and 100\*(1-α)% confidence interval

For each of n subjects  $t_j$  (j=1,...,n) specifies the exposure time. The number of occurrences of a treatment emergent event will be modeled to follow approximately a Poisson process with

constant intensity  $\theta$ . The rate parameter  $\theta$  will be estimated as  $\lambda = D/T$ , where  $T = \sum_{i=1}^{n} t_{j}$  and D

is the number of events (episodes). Conditionally on T, an exact  $100*(1-\alpha)\%$  confidence interval for a Poisson variable with parameter  $\theta T$  and observed value D can be obtained based on

(Garwood, 1936), from which an exact  $100*(1-\alpha)\%$  confidence interval for D/T will be derived as follows (Sahai, 1993; Ulm, 1990):

Lower confidence limit  $L = \frac{0.5c_{\alpha/2,2D}}{T}$  for D>0, 0 otherwise,

Upper confidence limit 
$$U = \frac{0.5c_{1-\alpha/2,2D+2}}{T}$$

where  $c_{\alpha k}$  is the  $\alpha$  th quantile of the Chi-square distribution with k degrees of freedom.

# 5.5 Rule of exclusion criteria of analysis sets

Protocol deviations for exclusion from analysis sets are defined in Table 5-1.

Table 5-1 Subject classification rules

| Analysis set | PD Categories Codes that cause subject to be excluded | Non-PD criteria that cause a subject to be excluded |
|---|---|---|
| Randomization set | NA | Misrandomized subject |
| FAS (Full Analysis Set) | DVSPID: INCL02; OTH30 | Misrandomized subject |
| Safety | DVSPID: INCL02; OTH30 | Subjects who did not take any study treatment |

INCL02: ICF missing or not signed prior to initiating study procedure

OTH30: Severe ICH-GCP non-compliance of study site

# 5.6 Clinician reported outcomes

# 5.6.1 Usability and hazard assessment of the 2 mL pre-filled syringe

The goal is to measure and evaluate the usability of the 2mL pre-filled syringe during observed use. During the first 2mL self-injection at the respective visits (Randomization and Week 1), site staff will observe and complete the self-injection assessment checklist (Table 5-2) to assess the ability to follow the instructions for use (IFU). The possible hazard checklist (Table 5-3) will be assessed for the 2mL self-injection at each of the two visits.

Primary usability assessment:

• Assessment of successful self-administration by the subject at Week 1. Successful self-injection is achieved when the subject performs all required steps effectively and safely to deliver the correct dose from the device at the correct injection site. The sequence of user steps (as per IFU) that are minimally required are P8, P10, P11, P12, P13, P14 (Table 5-2), these 6 critical steps will be used to define successful administration. The general passing usability goal for 'successful use' task completion will be defined as ≥ 90% pass rate following these steps.

Secondary usability assessment:

- Assessment of subject use errors that occur during the First Use at Randomization (after initial training) and repeated self-injection at Week 1 (without retraining).
- Assessment of successful First Use by subject after initial training (at Randomization), for subjects who successfully perform the self-injection as defined above for the primary usability assessment (i.e. P8, P10, P11, P12, P13, P14).

Table 5-2 Self injection assessment checklist (pre-filled syringe)

| No. | Instruction for use (IFU) indicated steps | Required for successful administration |
|---|---|---|
| P1 | Washed hands with soap and water | No |
| P2 | Cleaned the injection site | No |
| P3 | Removed the safety syringe from the outer box | No |
| P4 | Took syringe out of the tray | No |
| P5 | Checked expiration date on syringe label | No |
| P6 | Inspected the safety syringe for damage | No |
| P7 | Inspected liquid for brown discoloration or particles | No |
| P8 | Removed needle cap from safety syringe | Yes |
| P9 | Discarded needle cap | No |
| P10 | Pinched the skin at injection site | Yes |
| P11 | Inserted the needle into skin | Yes |
| P12 | Held onto the finger flange | Yes |
| P13 | Fully depressed plunger until end point | Yes |
| P14 | Held plunger pressed fully down and syringe in place for 5 seconds | Yes |
| P15 | Kept plunger fully depressed while lifting the needle straight from injection site | No |
| P16 | Released the plunger | No |
| P17 | Allowed syringe guard to automatically activate and cover the needle | No |
| P18 | Disposed used safety syringe in a sharps container | No |

#### Table 5-3 Possible hazard assessment checklist

| No. | Possible hazard assessment checklist |
|---|---|
| H1 | Was there a needle stick in a critical area (e.g. eye, carotid artery)? |
| H2 | Was there a needle stick in a non-critical area?1 |
| H3 | Was any part of the device swallowed? If yes, please specify. |
| H4 | Was an immediate-type allergic reaction noticed to device material? |
| H5 | Was increased pain noticed by the patient due to a bent needle? |
| H6 | Was the breakage of the device observed? <sup>2</sup> |
| H7 | Was swallowing of material debris observed? <sup>3</sup> |
| H8 | Was any other problem observed? <sup>3</sup> |
| H9 | Was less than the full dose administered? <sup>4</sup> |

# 5.7 Patient reported outcomes

The impact of psoriasis on various aspects of subjects' health-related quality of life will be assessed by the following instruments in this trial:

- DLQI
- •

# 5.7.1 Dermatology Life Quality Index (DLQI)

The DLQI is a 10-item general dermatology disability index designed to assess Health-related quality of life in adult subjects with skin diseases (e.g. psoriasis). The measure is self-administered and includes six domains of symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment.

The scoring of each question is as follows:

- Very much: Scored 3
- A lot: Scored 2
- A little: Scored 1
- Not at all: Scored 0
- Not relevant: Scored 0
- Question unanswered: Scored 0
- Question 7: "prevented work or studying": Scored 3

The DLQI total score will be calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more Quality of Life is impaired.

Meaning of DLQI Scores:

- 0-1= no effect at all on subject's life
- 2-5= small effect on subject's life
- 6-10= moderate effect on subject's life
- 11-20= very large effect on subject's life
- 21-30= extremely large effect on subject's life

<sup>&</sup>lt;sup>1</sup> Excluding the actual injection into the appropriate injection site of the body

<sup>&</sup>lt;sup>2</sup> If yes, then it is to be specified under which circumstances breakage occurred and which parts were affected, as well any additional problems (e.g. injuries) due to the breakage are to be described.

<sup>&</sup>lt;sup>3</sup> If yes, then it is to be specified. Possible events might include: irritated skin; drug too cold when injected; the drug or device upon visual inspection appeared unsuitable for injection; intradermal instead of subcutaneous injection; and other events.

<sup>&</sup>lt;sup>4</sup> If yes, then it is to be specified why, e.g. leakage from injection site, early removal.

The DLQI will be analyzed under six headings as follows:

- Symptoms and feelings: questions 1 and 2, score maximum 6
- Daily activities: questions 3 and 4, score maximum 6
- Leisure: questions 5 and 6, score maximum 6
- Work and school: question 7, score maximum 3
- Personal relationships: questions 8 and 9: score maximum 6
- Treatment: question 10, score maximum 3

Interpretation of incorrectly completed questionnaires:

There is a very high success rate of accurate completion of the DLQI. However, sometimes subjects do make mistakes.

- 1. If one question is left unanswered this is scored 0.
- 2. If two or more questions are left unanswered the questionnaire will not be scored.
- 3. If question 7 is answered 'yes' this will be scored 3. If question 7 will be answered 'no' or 'not relevant' but then either 'a lot' or 'a little' is ticked this will then be scored 2 or 1, respectively.
- 4. If two or more response options are ticked, the response option with the highest score will be recorded.
- 5. If there is a response between two tick boxes, the lower of the two score options will be recorded.
- 6. If one item is missing from a two- item subscale that subscale will not be scored.

Handling of missing values:

- If there is only one missing score per visit, it will be imputed with 0, and then the subscale including this item and the total score are derived accordingly.
- If there are two or more missing scores per visit, LOCF will be applied to the individual question scores, subscale scores, and total score, separately (i.e. LOCF is NOT applied to the 10 individual question scores for further derivation of the 6 subscale scores and 1 total score).

Of note, in situations where subjects responded to more questions than what was expected or required, the "most severe" answer was entered into the WriteResult (vendor for PRO data) database. In most cases the Self-Evident Corrections (SECs) were defined correctly, however, the SEC regarding question 7A/7B was not designed to select the "most severe" answer. This was confirmed with Novartis HEOR and communicated to the AIN team.





# 5.7.3 Self-injection Assessment Questionnaire (SIAQ)

The Self-Injection Assessment Questionnaire (SIAQ) is a questionnaire to measure overall subject experience with subcutaneous self-injection, and to investigate its psychometric properties. The SIAQ is composed of two modules: the PRE-module and the POST-module. The PRE-module, which is completed at Randomization before the first self-injection (baseline), includes 7 items grouped into three domains: feelings about injections, self-confidence and satisfaction with self-injection. The POST-module, which is completed following the two self-injections, includes several items addressing five principal domains: feelings about injections, self-confidence, injection-site reactions, ease of use, satisfaction plus a single item assessing self-image. Subjects will rate each item of the SIAQ on a 5-point semantic Likert-type scale ranging from 1 (worst experience) to 5 (best experience). Item score will be transformed to obtain a score ranging from 0 (worst experience) to 10 (best experience). The domain score will then be calculated as the mean of the item scores included in the domain.

Respondent rates each item of the PRE SIAQ and items 1-9 and 15-21 of the POST SIAQ on a 5-point semantic Likert-type scale, and items 10-14 of the POST SIAQ on a 6-point semantic Likert-type scale. For all items, a score of 1 corresponds to the subject's worst experience and a score of 5 or 6 corresponds to the subject's best experience.

The scoring of domains is performed in 2 steps:

- 1. The raw item scores ranging from 1 to 5 are transformed into scores ranging from 0 (worst experience) to 10 (best experience).
- 2. The transformed scores for items contributing to a domain are then averaged into a domain score (Table 5-5).

Table 5-5 Scoring of domains from raw item scores

| | Items | Transformed item score | Domain score calculation | Domain score range |
|---|---|---|---|---|
| PRE-module domain | | | | |
| FL | 1-3 | ((raw score)-1)*2.5 | Average of transformed item scores | 0-10 |
| CO | 4-6 | ((raw score)-1)*2.5 | | |
| SA | 7 | ((raw score)-1)*2.5 | | |
| POST- module domain | | | | |

| FL | 1-3 | ((raw score)-1)*2.5 | Average of transformed item scores | 0-10 |
|----|-------|---------------------|------------------------------------|------|
| IM | 4 | ((raw score)-1)*2.5 | | |
| CO | 5-7 | ((raw score)-1)*2.5 | | |
| RE | 8-9 | ((raw score)-1)*2.5 | | |
| EU | 10-14 | ((raw score)-1)*2 | | |
| SA | 15-21 | ((raw score)-1)*2.5 | | |

FL=Feeling about injection, IM=Self-Image, CO=Self-Confidence, RE=Pain and skin reaction during or after the injection, EU=Ease of use of the self-injection device, SA=Satisfaction with Self-injection

#### PRE-module:

- Item 1= In general, how afraid are you of needles?;
- Item 2= In general, how afraid are you of having an injection?;
- Item 3= How anxious do you feel about giving yourself an injection?;
- Item 4= How confident are you about giving yourself an injection in the right way?;
- Item 5= How confident are you about giving yourself an injection in a clean and sterile way?;
- Item 6= How confident are you about giving yourself an injection safely?;
- Item 7= Overall, how satisfied are you with your current way of taking your medication (self-injection)?

#### POST-module:

- Item 1= In general, how afraid are you of needles?;
- Item 2= In general, how afraid are you of having an injection?;
- Item 3= How anxious do you feel about giving yourself an injection?;
- Item 4= How embarrassed would you feel if someone saw you with the self-injection device?;
- Item 5= How confident are you about giving yourself an injection in the right way?;
- Item 6= How confident are you about giving yourself an injection in a clean and sterile way?;
- Item 7= How confident are you about giving yourself an injection safely?;
- Item 8a= During and/or after the injection, how bothered were you by: pain";
- Item 8b= During and/or after the injection, how bothered were you by: burning sensation";
- Item 8c= During and/or after the injection, how bothered were you by: cold sensation";
- Item 9a= During and/or after the injection, how bothered were you by: itching at the injection site?";
- Item 9b= During and/or after the injection, how bothered were you by: redness at the injection site?";
- Item 9c= During and/or after the injection, how bothered were you by: swelling at the injection site?";
- Item 9d= During and/or after the injection, how bothered were you by: bruising at the injection site?";
- Item 9e= During and/or after the injection, how bothered were you by: hardening at the injection site?";
- Item 10= How difficult or easy was it to remove the cap?;
- Item 11= How difficult or easy was it to depress the device?;
- Item 12= How difficult or easy was it to administer the injection without any help?;
- Item 13= How difficult or easy was it to use the self-injection device?;
- Item 14= How does the device fit in your hand?;
- Item 15= How easy was it to give yourself an injection?;
- Item 16= How satisfied are you with how often you give yourself an injection?;
- Item 17= How satisfied are you with the time it takes to inject the medication?;
- Item 18= Overall, how satisfied are you with your current way of taking your medication (self-injection)?:
- Item 19= Overall, how convenient is the self-injection device?;
- Item 20= After this study, would you choose to continue self-injecting your medication?;
- Item 21= After this study, how confident would you be to give yourself injections at home?



Alberti KGMM, Eckel RH, Grundy SM, et al (2009) Harmonizing the metabolic syndrome: a joint interim statement of the international diabetes federation task force on epidemiology and prevention; national heart, lung, and blood institute; american heart association; world heart federation; international atherosclerosis society; and international association for the study of obesity. Circulation; 120: 1640-1645.

Bishop YMM, Fienberg SE, Holland PW (1991) Discrete multivariate analysis. Cambridge MA, 11<sup>th</sup> ed. The MIT Press

Bretz F, Maurer W, Brannath W, Posch M (2009) A graphical approach to sequentially rejective multiple test procedures. Statistics in Medicine; 28: 586-604.

'CIS liver safety' guidance, available in Cabinets/CREDI TABULU/B&SR/CIS Process Documentation/Guidances (outside of ESOPS)/Others

Clopper CJ, Pearson ES (1934). The use of confidence or fiducial limits illustrated in the case of the binomial. Biometrika, 26; 404–413.



Fredriksson T, Pettersson U (1978) Severe psoriasis—oral therapy with a new retinoid. Dermatologica; 157:238–44.

Garwood, F (1936). Fiducial limits for the Poisson distribution. Biometrika, 46; 441–453.

Gottlieb A, Griffiths CEM, Ho VC, et al (2005) Efficacy and tolerability of oral pimecrolimus in the treatment of moderate to severe chronic plaque type psoriasis: a double-blind, multicentre, randomized dose-finding trial. Br J Dermatol; 152:1219-27.

Kenward, M. and Roger, J. (1997). Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. Biometrics; 53: 983-997.

Lachin JM (2000) The assessment of relative risks . New York: Wiley

Little, R.J.A and Rubin, D.B. (2002). Statistical Analysis with Missing Data. Wiley Series in Probability and Statistics, Chapter 10.

Menter A, Gottlieb A, Feldman S, et al (2008) Guidelines of care for the management of psoriasis and psoriatic arthritis – Section 1. Overview of psoriasis and guidelines of care for the treatment of psoriasis with biologics. J Am Acad Dermatol; 58:826-850.

Newcombe RG (1998) Two-sided confidence intervals for the single proportion: comparison of seven methods. Statistics in Medicine; 17: 857-872.

Papp KA, Tyring S, Lahfa M et al (2005) A global phase II randomized controlled trial of etanercept in psoriasis: safety, efficacy, and effect of dose reduction. Br J Dermatol; 152:1304-12.

Rubin, D.B. (1987). Multiple Imputation for Nonresponse in Surveys. New York: Wiley.

Sahai H, Khurshid Anwer (1993). Confidence intervals for the mean of a poisson distribution: a review. Biom J, 35 (7); 857-867

Sampson HA, Muñoz-Furlong A, Bock SA, et al (2005) Symposium on the Definition and Management of Anaphylaxis: Summary report. J Allergy Clin Immunol 2005;115:584-91.

Sampson HA, Muñoz-Furlong A, Campbell RL, et al (2006) Second Symposium on the Definition and Management of Anaphylaxis: Summary Report - Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network Symposium. Ann Emerg Med;47(4):373-80.

Schaefer, J.L. (1997). Analysis of Incomplete Multivariate Data, Chapman&Hall.

Ulm K (1990). A simple method to calculate the confidence interval of a standard mortality ratio. American Journal of Epidemiology, 131(2); 373-375

Weisman S, Pollack CR, Gottschalk RW (2003) Psoriasis disease severity measures: comparing efficacy of treatments for severe psoriasis. J Dermatology Treat; 14: 158-165.